

### Statistical Analysis Plan

NCT Number: NCT03710486

Title: Vedolizumab and anti-TNFs Outcomes in Real-World Biologic Ulcerative

Colitis and Crohn's Disease Patients (EVOLVE) – IBERIA

Study Number: Vedolizumab-5047

Document Version and Date: 6.0, 17FEB2022

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

| Trial Name: | EVOLVE study |
|---|---|
| Trial Title: | Vedolizumab and anti-TNFs Outcomes in Real-World Biologic Ulcerative Colitis and Crohn's Disease Patients (EVOLVE) – IBERIA |
| Protocol No.: | TAK-VEZ-2018-01 |
| Sponsor: | Takeda Farmacéutica España SA |

| Reference to version and date of protocol and SAP on which report is based | |
|---|---|
| Protocol version: | 2.0 |
| Protocol date: | 23MAY2019 |
| SAP Version: | NA ONE |
| SAP date: | NA SS |

| Date: | 17FEB2022 |
|----------|-----------|
| Version: | 6.0 |

Performed by:

Performed for:

Takeda

Property



## 1. Approvals (signatures)

The signatures on this page indicate the review and approval of the statistical analysis plan of the EVOLVE study.





Study : EVOLVE

Version : 6.0

Date : 17FEB2022

### Index

| 1. | Approvals (signatures) | 2 |
|---|---|---|
| 2. | Distribution List | 14 |
| 3. | Document Version History | 14 |
| 4. | Study objectives | 15 |
| 4.1 | Primary objective | 15 |
| 4.2 | | |
| 4.3 | Secondary objectives Exploratory Objectives Overall study design Study design | 15 |
| 5. | Overall study design | 15 |
| 5.1 | Study design | 15 |
| 5.2 | Sample size | 16 |
| | Cample size | 10 |
| 5.3 | Sample size Changes to the protocol General statistical considerations | 16 |
| 6. | General statistical considerations | 16 |
| 6.1 | Study population | 16 |
| 6.2 | General statistical considerations Study population General issues Presentation/Format of the results | 16 |
| 6.3 | Presentation/Format of the results | 17 |
| 6.4 | Level of significance and multiplicity | 17 |
| 6.5 | Handling of dropouts and missing data | 17 |
| 7. | Description of the statistical analysis | 17 |
| 7.1 | Definitions of variables | |
| 7.2 | Hypothesis and statistical methods | 23 |
| | 7.2.1 Univariate analysis. Descriptive statistics | 23 |
| | 7.2.2 Bivariate analysis | 23 |
| 7.3 | Demographic and baseline characteristics | 24 |
| 7.4 | Primary objective analysis | 24 |
| ) | 7.4.1 Descriptive analysis | 24 |
| | 7.4.2 Endpoint analysis | 24 |
| 7.5 | Analysis of secondary objectives | |
| 7.6 | Exploratory Objectives | 31 |
| 8. | References | 32 |



Study : EVOLVE

Date : 17FEB2022


| 9. | Results3 | | |
|-----|----------|---------------------------------------------------|------|
| 9.1 | Stud | . 33 | |
| 9.2 | Des | criptive analysis | .35 |
| | 9.2.1 | Groups description | . 35 |
| | 9.2.2 | By treatment | . 39 |
| | 9.2.3 | By treatment (CD patients) | . 60 |
| | 9.2.4 | By treatment line (CD-VDZ patients) | . 60 |
| | 9.2.5 | By treatment line (CD-Other Biologic Patients) | |
| | 9.2.6 | By treatment (UC patients) | |
| | 9.2.7 | By treatment line (UC-VDZ patients) | . 62 |
| | 9.2.8 | By treatment line (UC-Other Biologic Patients) | . 62 |
| 9.3 | Prim | pary Objective (Descriptive analysis) | . 63 |
| | 9.3.1 | Descriptive by treatment | . 63 |
| | 9.3.2 | By treatment (CD patients) | . 70 |
| | 9.3.3 | By treatment line (CD-VDZ patients) | |
| | 9.3.4 | By treatment line (CD-Other Biologic Patients) | |
| | 9.3.5 | By treatment (UC patients) | |
| | 9.3.6 | By treatment line (UC-VDZ patients) | |
| | 9.3.7 | By treatment line (UC-Other Biologic Patients) | |
| 9.4 | | pary objective (Endpoint analysis) | |
| | 9.4.1 | PS-IPTW. | 73 |
| | 9.4.1 | Discontinuation | |
| | 9.4.2 | Time to treatment discontinuation | |
| | 9.4.4 | Duration of treatment | |
| | 9.4.5 | Intensification | |
| 1 | 0. | Time to first intensification | |
| Č | 9.4.6 | | |
| | 9.4.7 | Clinical response | |
| | 9.4.8 | Clinical remission | |
| | 9.4.9 | Endoscopic response at 52 weeks | |
| | 9.4.10 | Endoscopic remission at 52 weeks | |
| | 9.4.11 | Biochemical remission based on CRP | 168 |
| | 9.4.12 | Biochemical remission based on fecal calprotectin | 168 |



Table 2.2.8

**Table 2.2.9** 

Table 2.2.10

**Table 2.2.11** 

**Table 2.2.12** 

**Table 2.3.1** 

**Table 2.4.1** 

**Table 2.5.1** 

#### STATISTICAL ANALYSIS PLAN

Study: EVOLVE

Version: 6.0 Date: 17FEB2022

| 9.5 | Sec | ondary objectives |
|---|---|---|
| | | Describe the real world clinical effectiveness of VDZ vs. other biologics at least hs post-treatment initiation (in a subgroup of patients with adequate follow-up) |
| | | Quantify healthcare resource utilization including the rates of healthcare and (HCP) and emergency department (ED) visits, hospitalizations and atory Bowel Disease (IBD) related surgical procedures |
| | 9.5.3 | Identify predictors of response to VDZ |
| | index tre | Describe treatment patterns, clinical effectiveness and safety events for at least ction phase of the subsequent biologic regimen for patients who discontinue atment in the VDZ cohort and initiate a second -line biologic within 6 months ex treatment discontinuation |
| Table | 9.5.5<br>other bio | Describe the safety events occurring post biologic treatment initiation (VDZ or logics) |
| rabie | Index | and |
| Table | 1.1.1 | Patients recruited, valid and excluded33 |
| Table | 1.1.2 | Follow-up |
| Table | 2.1.1 | Groups and subgroups35 |
| Table | 2.2.1 | Demographics39 |
| Table | 2.2.2 | Disease Characteristics – CD patients |
| Table | 2.2.3 | Disease Activity – CD patients |
| Table | 2.2.4 | Disease Characteristics – UC patients |
| Table | 2.2.5 | Disease Activity – UC patients |
| Table | 2.2.6 | Diagnostic imaging 50 |
| Table | 2.2.7 | Laboratory determinations51 |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

Extra Intestinal Manifestations ...... 52

Comorbid medical conditions......54

Biologic treatment pre index treatment ...... 56

Non-biologic treatment...... 58

End of study ...... 59

Demographics (CD patients) ...... 60

Demographics (CD-VDZ patients)......60

Demographics (CD-Other Biologic patients)......61



Study : EVOLVE

Date : 17FEB2022


| <b>Table 2.6.1</b> | Demographics (UC patients) | 61 |
|---|---|---|
| <b>Table 2.7.1</b> | Demographics (UC-VDZ patients) | |
| <b>Table 2.8.1</b> | Demographics (UC-Other Biologic patients) | 62<br>63 |
| <b>Table 3.1.1</b> | Biologic index treatment I | 63 |
| <b>Table 3.1.2</b> | Biologic index treatment II | na . w / |
| <b>Table 3.1.3</b> | Follow-up | 68 |
| <b>Table 3.1.4</b> | Concomitant treatment | hu . |
| <b>Table 3.2.1</b> | Biologic index treatment I (CD patients) | 70 |
| <b>Table 3.3.1</b> | Biologic index treatment I (CD-VDZ patients) | 70 |
| <b>Table 3.4.1</b> | Biologic index treatment I (CD-Other Biologic patients) | 71 |
| <b>Table 3.5.1</b> | Biologic index treatment I (UC patients) | 71 |
| <b>Table 3.6.1</b> | Biologic index treatment I (UC-VDZ patients) | 72 |
| <b>Table 3.7.1</b> | Biologic index treatment I (UC-Other Biologic patients) | 72 |
| Table 4.1.1 | Descriptive analysis pre and post PS-IPTW (CD patients) | 73 |
| <b>Table 4.1.2</b> | Descriptive analysis pre and post PS-IPTW (UC patients) | 76 |
| <b>Table 4.1.3</b> | Descriptive analysis pre and post PS-IPTW (CD patients – First line) | 79 |
| <b>Table 4.1.4</b> | Descriptive analysis pre and post PS-IPTW (UC patients – First line) | 82 |
| <b>Table 4.1.5</b> | Descriptive analysis pre and post PS-IPTW (CD patients – Second line) | 85 |
| <b>Table 4.1.6</b> | Descriptive analysis pre and post PS-IPTW (UC patients – Second line) | 88 |
| <b>Table 4.2.1</b> | Discontinuation | 91 |
| Table 4.2.2 values) | CD patients with VDZ - Discontinuation Logistic regression model () | 0- |
| Table 4.2.3 (estimated Q | CD patients with VDZ – Discontinuation Logistic regression mod | |
| Table 4.2.4 values | UC patients with VDZ – Discontinuation Logistic regression model () | |
| Table 4.2.5 | UC patients with VDZ - Discontinuation Logistic regression mod | |
| (estimated O | R)1 | |
| Table 4.2.6<br>model (p-valu | CD patients with Other Biologic – Discontinuation Logistic regressions: | |
| Table 4.2.7 model (estim | CD patients with Other Biologic – Discontinuation Logistic regression ated OR) | |
| Table 4.2.8 | UC patients with Other Biologic – Discontinuation Logistic regressions: | n |



Study : EVOLVE


Date: 17FEB2022

| • | Biologic – Discontinuation Logistic regression |
|---|---|
| Table 4.3.1 Time to treatment disco | ntinuation (Months) 108 |
| Table 4.4.1 Duration of treatment (M | Ionths) |
| | A-2 |
| Table 4.5.2 CD patients with VDZ - model (p-values) | - One intensification or more Logistic regression 133 |
| • | - One intensification or more Logistic regression |
| | - One intensification or more Logistic regression |
| Table 4.5.5 UC patients with VDZ - | - One intensification or more Logistic regression |
| regression model (n-values) | 137 |
| Table 4.5.7 CD patients with Other regression model (estimated OR) | Biologic – One intensification or more Logistic |
| | Biologic – One intensification or more Logistic |
| | Biologic – One intensification or more Logistic |
| Table 4.6.1 Time to first intensification | ion (Months) 141 |
| Table 4.7.1 Clinical response at 14 v | veeks148 |
| Table 4.7.2 Clinical response at 52 v | veeks156 |
| | Clinical response at 52 weeks Logistic regression |
| | Clinical response at 52 weeks Logistic regression |
| · · | Clinical response at 52 weeks Logistic regression |
| | Clinical response at 52 weeks Logistic regression |
| | Biologic – Clinical response at 52 weeks Logistic |
| <u>-</u> | Biologic – Clinical response at 52 weeks Logistic |



Study : EVOLVE


Date: 17FEB2022

| Table 4.7.9 UC patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (p-values) |
|---|
| Table 4.7.10 UC patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (estimated OR) |
| Table 4.8.1 Clinical remission at 14 weeks |
| Table 4.8.2 Clinical remission at 52 weeks |
| Table 4.8.3 CD patients with VDZ – Clinical remission at 52 weeks Logistic regression model (p-values) |
| Table 4.8.4 CD patients with VDZ – Clinical remission at 52 weeks Logistic regression model (estimated OR) |
| Table 4.8.5 UC patients with VDZ – Clinical remission at 52 weeks Logistic regression model (p-values) |
| Table 4.8.6 UC patients with VDZ – Clinical remission at 52 weeks Logistic regression model (estimated OR) |
| Table 4.8.7 CD patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (p-values) |
| Table 4.8.8 CD patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (estimated OR) |
| Table 4.8.9 UC patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (p-values) |
| Table 4.8.10 UC patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (estimated OR) |
| Table 4.9.1 Endoscopic esponse at 52 weeks |
| Table 4.9.2 CD patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (p-values) |
| Table 4.9.3 CD patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (estimated OR) |
| Table 4.9.4 UC patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (p-values) |
| Table 4.9.5 UC patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (estimated OR) |
| Table 4.9.6 CD patients with Other Biologic – Endoscopic response at 52 weeks Logistic regression model (p-values) |
| Table 4.9.7 CD patients with Other Biologic – Endoscopic response at 52 weeks Logistic regression model (estimated OR) |



Study : EVOLVE


Date : 17FEB2022

| Table 4.9.8<br>Logistic regr | UC patients with Other Biologic – Endoscopic response at 52 weeks ession model (p-values) |
|---|---|
| Table 4.9.9<br>Logistic regr | UC patients with Other Biologic – Endoscopic response at 52 weeks ession model (estimated OR) |
| Table 4.10.1 | Endoscopic remission at 52 weeks167 |
| Table 4.11.1 | Biochemical remission based on CRP at 14 weeks 168 |
| Table 4.11.2 | Biochemical remission based on CRP at 52 weeks168 |
| Table 4.12.1 | Biochemical remission based on fecal calprotectin at 14 weeks 168 |
| Table 4.12.2 | Biochemical remission based on fecal calprotectin at 52 weeks 168 |
| Table 5.2.1 | Health resource utilization – CD with VDZ patients |
| <b>Table 5.2.2</b> | Health resource utilization related to the pathology – CD with VDZ patients173 |
| <b>Table 5.2.3</b> | Health resource utilization – CD patients with other biologic 177 |
| Table 5.2.4 other biologi | Health resource utilization related to the pathology – CD patients with c |
| Table 5.2.1 | Health resource utilization – UC patients with VDZ184 |
| <b>Table 5.2.2</b> | Health resource utilization related to the pathology – UC patients with VDZ184 |
| <b>Table 5.2.3</b> | Health resource utilization – CD patients with other biologic 184 |
| <b>Table 5.2.4</b> | Health resource utilization related to the pathology – UC patients with |
| other biologi | c184 |
| Table 5.4.1 | Patients who discontinue index treatment in the VDZ cohort and initiate a |
| | piologic within 6 months post-index treatment discontinuation 186 |
| Table 5.4.1 | New treatment |
| Table 5.4.2 | Posology (mg) by treatment |
| Table 5.4.1 | New treatment – Response and remission 14 weeks 189 |
| <i>\( \dots \)</i> | New treatment – Adverse Events 190 |
| Table 5.5.1 | Adverse Events |
| Table 5.5.2 | Adverse event (incidence)194 |
| <b>T</b> able 5.5.3 | Serious Adverse event (incidence)195 |
| Table 5.5.4 | Related with treatmetn Adverse Event (incidence)195 |
| Table 5.5.5 | Related with treatment Serious Adverse Event (incidence) 195 |
| Table 5.5.6 (incidence) | Adverse event - Infections, serious infections and malignancies 195 |
| Table 5.5.1 | Adverse event (incidence rate) |
| <b>Table 5.5.2</b> | Serious Adverse event (incidence rate)196 |



Study : EVOLVE

Date : 17FEB2022


| Table 5.5.3 | Related with index date Adverse Event (incidence rate) | 197 |
|---|---|---|
| <b>Table 5.5.4</b> | Related with index date Serious Adverse Event (incidence rate) | |
| Table 5.5.5 (incidence ra | Adverse event - Infections, serious infections and malignanci | 19 |
| <b>Table 5.5.6</b> | Adverse Events I – CD patients with VDZ | 198 |
| Table 5.5.7 | Adverse Events II – CD patients with VDZ | 199 |
| <b>Table 5.5.8</b> | Adverse Events III – CD nationts with VD7 | 200 |
| <b>Table 5.5.9</b> | Adverse Events I – CD patients with Other Biologic | 201 |
| Table 5.5.10 | Adverse Events II – CD patients with Other Biologic | 202 |
| Table 5.5.11 | Adverse Events III – CD patients with Other Biologic | 203 |
| Table 5.5.12 | Adverse Events II – CD patients with Other Biologic | 204 |
| Table 5.5.13 | Adverse Events II – UC patients with VDZ | 204 |
| Table 5.5.14 | Adverse Events III – UC patients with VDZ | 204 |
| Table 5.5.15 | Adverse Events I – UC patients with Other Biologic | 204 |
| Table 5.5.16 | Adverse Events II – UC patients with Other Biologic | 204 |
| Table 5.5.17 | Adverse Events III – UC patients with Other Biologic | 204 |
| Figure index | | |
| Figure 4.1.1 | Density Plot – pre PS-IPTW (CD) | 75 |
| Figure 4.1.2 | Density Plot Post-IPTW (CD) | |
| Figure 4.1.3 | Love Plot (CD) | |
| Figure 4.1.4 | Box Plots (CD) | |
| Figure 4.1.5 | Density Plot – pre PS-IPTW (UC) | |
| Figure 4.1.6 | Density Plot – Post-IPTW (UC) | |
| Figure 4.1.7 | Love Plot (UC) | 78 |
| Figure 4.1.8 | Box Plots (UC) | . 78 |
| Figure 4.1.9 | Density Plot – pre PS-IPTW (CD – First line) | 81 |
| Figure 4.1.10 | Density Plot – Post-IPTW (CD – First line) | 81 |
| Figure 4.1.11 | Love Plot (CD – First line) | 81 |
| Figure 4.1.12 | Box Plots (CD – First line) | 81 |
| Figure 4.1.13 | | |
| | Density Plot - pre PS-IPTW (UC - First line) | . 84 |



Study: EVOLVE Version: 6.0

Date: 17FEB2022

Love Plot (UC - First line)......84 Figure 4.1.15 Figure 4.1.16 Box Plots (UC - First line) ...... 84 Figure 4.1.17 Figure 4.1.18 Figure 4.1.19 Figure 4.1.20 Figure 4.1.21 Density Plot - Post-IPTW (UC - Second line)......90 Figure 4.1.22 Figure 4.1.23 Love Plot (UC - Second line)..... Property of Takeda: For Non-Commercial Use Only and Subject in Box Plots (UC – Second line) ...... 90 Figure 4.1.24




Date: 17FEB2022

#### **ABBREVIATIONS AND DEFINITIONS**

5-ASA 5-aminosalicylic acid

ΑE Adverse Event

**AIDS** Acquired immune deficiency syndrome

ALT Alanine transaminase ANOVA Analysis of variance **AST** Aspartate transaminase

BMI **Body Mass Index** BUN Blood urea nitrogen CD Crohn's disease

CHF Congestive heart failure Confidence interval CI CKD Chronic kidney disease

**CPPD** Calcium pyrophosphate dihydrate

**CVA** Cerebrovascular accident ED **Emergency Department** 

and Subject to the Applicable Terms of Use and Subject to the Applicable Terms of Use Good Pharmacoepidemiology Practices **GPP** 

Healthcare professional **HCP** Harvey-Bradshaw Index HBI Inflammatory bowel disease **IBD** 

Inverse Probability Treatment Weighting **PS-IPTW** Medical Dictionary for regulatory activities MedDRA

Magnetic resonance imaging MRI

NA Not applied OR Odds Ratio RR Relative Risk

C Reactive Protein

**PSC** Primary sclerosing colangitis

Preferred Term

**Q**1/Q3 First and third quartile

SES-CD Simple endoscopic score for Crohn's disease

SAS Statistical Analysis Software

SD Standard Deviation SOC System Organ Class

TIA Transient ischemic attack

UC Ulcerative colitis



VDZ Vedolizumab

Properly of Takeda: For Mon. Commercial Use Only and Subject to the Applicable Terms of Use



### 2. Distribution List

| 2. Distribution List | | |
|-----------------------------|-----------------|----------------|
| Name | Function / Role | Office/Sponsor |
| | Sponsor | Takeda |
| | Sponsor | Takeda |
| | Sponsor | Takeda |
| | Sponsor | Takeda |
| | Sponsor | Takeda |
| 3. Document Version History | | |

# 3. Document Version History

| Version | Effective Date | Significant Changes |
|---|---|---|
| 1.0 | 27MAY2020 | New endpoints and Propensity score PS-IPTW methodology. |
| 2.0 | 15DEC2020 | A logistic regression with Other Biologic patients, all Kaplan-Meier's graphs and other minor changes. |
| 3.0 SON | 13JAN2021 | Additional covariates for PS-IPTW. Boxplots for analysis of the distribution of covariates after PS-IPTW. Other minor changes. |
| 4.0 | 24JAN2021 | Removed comments. |
| 5.0 | 03FEB2022 | Correct minor errors. |



| Study: EVOLVE |
|---------------|

Date: 17FEB2022

### 4. Study objectives

### 4.1 Primary objective

- Describe treatment patterns associated with first-line and second line biologic use (VDZ or other biologic: infliximab, adalimumab, or golimumab, [UC only]) (e.g., dose escalation, treatment discontinuation, and switching).
- Describe the real-world clinical effectiveness of the use (first-line and second line) VDZ vs. other biologics at least 6 months post-treatment initiation.

### 4.2 Secondary objectives

- Characterize patients treated with VDZ or other biologics (infliximab, adalimumab, or golimumab [UC only]) as first and second line biologic therapy in terms of demographics, medical, and treatment histories.
- Describe the real world clinical effectiveness of VDZ vs. other biologics at least 12 months post-treatment initiation (in a subgroup of patients with adequate follow-up available).
- Describe the safety events occurring post biologic treatment initiation (VDZ or other biologics).
- Quantify healthcare resource utilization including the rates of healthcare professional (HCP) and emergency department (ED) visits, hospitalizations and Inflammatory Bowel Disease (IBD) related surgical procedures.



# 5. Overall study design

### 5.1 Study design

This study is a 'non-interventional study' as defined in Directive 2001/20/EC and will follow the guidelines for GPP.

This means that:



| Study : EVOLVE |
|------------------|
| Date : 17FEB2022 |

- The assignment of a subject to a particular therapeutic strategy is not decided in advance by the study protocol but falls within current practice.
- No additional diagnostic or monitoring procedures shall be applied to the subjects.
- Epidemiological methods shall be used for the analysis of collected data.

The study is an ethics-approved, designed as a multicentre, retrospective cohort study of the medical charts of patients who were diagnosed with CD or UC and who initiated first- or second-line biologic treatment with VDZ or another biologic (infliximab, adalimumab, or golimumab [UC only]) (index event) during the eligibility period: January 2017 to date of site initiation.

The target sample size is approximately 400 patients (200 patients per treatment cohort: 1) VDZ and 2) other biologics. It is estimated that these patients will be included from across ~25 sites (20 in Spain and 5 in Portugal), resulting on average in ~8 patients per treatment cohort/site. The medical charts of patients with UC or CD who initiated first-line or second-line biologic treatment with VDZ or another biologic (infliximab, adalimumab, or golimumab [UC only]) during the eligibility period will be identified for potential enrolment.

### 5.2 Sample size

The primary objective of the study is descriptive. Therefore, the sample size calculation is based in the precision of a confidence interval estimation of a proportion. The study will recruit two types of patients; the distribution will be 1:1. Both groups will be evaluated separately in consequence we calculated a sample size calculation for each group.

We assumed the scenario of maximum indetermination (i.e., an expected proportion of 50%). To obtain a confidence interval of 95% of this proportion with a precision of 7.5% is necessary to recruit 171 patients. We expect a 10% of non-valid data so we will recruit 200 patients per group (400 patients in total).

- 200 patients treated with a first-line or second-line VDZ.
- 200 patients treated with first-line or second-line of other biologics (infliximab, adalimumab, golimumab).

### 5.3 Changes to the protocol

NÁ

### 6. General statistical considerations

### 6.1 Study population

Valid sample: Patients that meet all the inclusion criteria and none of exclusion.

#### 6.2 General issues



| Study : EVOLVE |
|------------------|
| Date : 17FEB2022 |

The content of the clinical database will be transferred to SAS® datasets for statistical analysis. All statistical analyses will be performed using the statistical package SAS® system insofuse version 9.4 or posterior.

In section 9 the tables of the statistical analysis are shown.

#### 6.3 Presentation/Format of the results

In general, for the continuous variables, the description of the mean, median and standard deviation is presented with an additional decimal and for the minimum and maximum values it is presented with the same level of accuracy as the raw data.

For the categorical variables, the percentages are presented with a decimal figure,

#### 6.4 Level of significance and multiplicity

The level of significance that will be adopted for all tests has been 0.05 bilateral.

No adjustment will be made for multiple comparisons or corrections for multiplicity.

#### Handling of dropouts and missing data 6.5

Missing data of PS-IPTW model variables will be imputed by means of PROC MI and FCS option (SAS software version 9.4 or posterior). Multiple imputation will include 25 datasets.

# 7. Description of the statistical analysis

#### 7.1 Definitions of variables

Index date: Date of the initiation of treatment (VDZ or other biologic)

Time of follow-up (months):

(Date of last time alive/Date of death - index date)/30.4375

Patients with follow-up of 12 months or more:

Patients with "Time of follow-up" equal or greater than 12: Yes

Patients without "Time of follow-up" equal or greater than 12: No

Time between index date and assessment (weeks):

(Date of assessment - Index date)/7

Time between intensification and index date (months):




Date: 17FEB2022

(Date of intensification – Date of index date)/30.4375

Time between induction and maintenance (weeks):

(Date of maintenance initial – date of induction initial)/7

Time between index treatment and new treatment (months):

(Date of new treatment initial - Index date)/30.4375

Number of visits (global and by type):

Sum of visits and sum of visit by type.

AEs duration (days):

(Date of resolution - Start of onset)+1

- Assessment for clinical response and remision:
- Subject to the Applicable Terms of Use site a o Select all assesments posterior to index date and with HBI value/Partial Mayo (CD or UC patients) or physician statuts other than missing, NA or Unknown.
  - o Select assesments inside time window 10-18 weeks for 14 weeks assessment and 46-58 weeks for 52 weeks assessment. For each patient the nearest assessment to 14 and 52 will be seleceted. In case of two evaluation at the same distance from 14 or 52 the latests assessment will be selected.
  - Patients without assessment inside time window:
    - If there is a discontinuation registred before 14 or 52 we will impute a "No" clinical remission and clinical response for 14 or 52 weeks assessment.
    - If there is not a discontinuation:
      - Select all assessments below time window (<10 weeks or <46</li> weeks). For each patient the latest assessment will be selected.

Assessment for clinical response and remission (New treatment):

ne same index date. The same methodology below for 14 weeks but using date of start of new treatment instead of

- Clinical response (CD patients):
  - o HBI score registered or calculated (if both are available used that registered in the clinical chart):
    - Yes:



Study: EVOLVE Version: 6.0 Date: 17FEB2022

- HBI score equal or less than 4: Clinical response = Yes.
- HBI score at index date equal or greater than 3:
  - o Reduction (difference from index date) equal or greater than 3: Clinical response = Yes.
  - plicable Terms of Use o Reduction (difference from index date) less than 3: Clinical response = No
- Other case: Physician assessment registered.
- No: Physician assessment registered
- Physician assessment registered:
  - Yes
- Remission or Partial remission: Clinical response = Yes o W
- Not in remission: Clinical response =No
- Unknown or NA: Missing
- No: Clinical response = Missing
- Clinical remission (CD patients):
  - o HBI score registered or calculated (if both are available used that registered in the clinical chart):
    - Yes:
- HBI score equal or less than 4: Clinical remission = Yes.
- HBI score greater than 4: Clinical remission = No
- No: Physician assessment registered.
- Physician assessment registered:
- Remission: Clinical remission = Yes
- Partial remission or not in remission Clinical remission =No
- Unknown or NA: Missing
- No: Clinical remission = Missing
- Clinical response (UC patients):
  - Partial Mayo score registered or calculated:
    - Yes:
- Partial Mayo score less than 4: Clinical response = Yes.
- Partial Mayo score at index date equal or greater than 2:
  - o Reduction (difference from index date) equal or greater than 2: Clinical response = Yes.



Study: EVOLVE Version: 6.0 Date: 17FEB2022

o Reduction (difference from index date) less than 2: Terms of Use Clinical response = No

- Other case: Physician assessment registered
- No: Physician assessment registered
- o Physician assessment registered:
  - Yes
- Remission or Partial remission: Clinical response = Yes
- Not in remission: Clinical response =No
- Unknown or NA: Missing
- No: Clinical response = Missing
- Clinical remission (UC patients):
  - o Partial Mayo score registered or calculated:
    - Yes:
- Partial Mayo score less than 2: Clinical remission = Yes.
- Partial Mayo score equal or greater than 2: Clinical remission =
- No: Physician assessment registered
- Physician assessment registered:
  - Yes
- Remission: Clinical remission = Yes
- Partial remission or not in remission: Clinical remission =No
- Unknown or NA: Missing
- No: Clinical remission = Missing
- Assessment for endoscopic response and remision:
  - Select all assesments posterior to index date and with SES-CD (only Cd patients) or endoscopic statuts other than missing, NA or Unknown.
  - Select assesments inside time window 28-76 weeks for 52 weeks assessment. For each patient the nearest assessment to 52 will be seleceted. In case of two evaluation at the same distance from 52 the latests assessment will be selected.
  - Patients without assessment inside time window: Select all assessments below time window <28 weeks. For each patient the latest assessment will be selected
- Endoscopic response at 52 weeks (CD and UC patients):
  - Endoscopy:



Study : EVOLVE


Date : 17FEB2022

- SES-CD score registered (only CD patients):
  - Yes
- SES-CD score equal or less than 2: Endoscopic response = Yes.
- SES-CD greater than 2 and SES-CD at index date equal 0: Endoscopic response = No.
- o In other case:
  - SES-CD at index date greater than 0 relative difference will be calculated {100\*(Index date – 52 weeks assessment)/Index date};
    - Greater or equal 50%: Endoscopic response=Yes
    - Less than 50: Endoscopic response=No
  - Other case: Endescopic response=Missing
- No: Physician assessment
- Physician assessment
  - Remission or Partial remission: Endoscopic response = Yes
  - Not in remission: Endoscopic response =No
- Endoscopic remission at 52 weeks (CD and UC patients):
  - o Endoscopy:
    - SES-CD score registered (only CD patients):
      - Yes
- SES-CD score equal or less than 2: Endoscopic remission = Yes.
- OSES-CD score greater than 2: Endoscopic remission = No
- No: Physician assessment
- Physician assessment:
  - Remission: Endoscopic remission = Yes
  - Partial remission or not in remission: Endoscopic remission =No
- Assessment for bioquimic remission based on CRP/fecal calcoprotectin at 14 and 52 weeks:
  - Select all assesments posterior to index date and with CRP/fecal calcoprotectin.
  - Select assessments inside time window >0-38 weeks for 14 weeks assessment and 28-76 weeks for 52 weeks assessment. For each patient the nearest assessment to 14 and 52 will be selected. In case of two evaluation at the same distance from 14 or 52 the latests assessment will be selected.




Date: 17FEB2022

- Biochemical remission based on CRP (CD and UC patients):
  - o CRP (mg/L):
    - <5: Biochemical remission = Yes</p>
    - >=5: Biochemical remission =No
- to the Applicable Terms of Use Biochemical remission based on fecal calprotectin (CD and UC patients):
  - Fecal calcoprotein (μg/g):
    - <250: Biochemical remission = Yes</p>
    - >=250: Biochemical remission =No
- Time to discontinuation (months):
  - o Is the treatment ongoing? = No
    - (date of discontinuation index date)/30.43
  - o Is the treatment ongoing? = Yes
    - Censured time: (date of the last assessment index date)/30.4375
- Time to first intensification (months):
  - o Is the treatment ongoing? = No
    - Has there been intensification? = Yes
      - (date of the first intensification index date)/30.4375
    - Has there been intensification? = No
      - Censured time: (date of discontinuation index date)/30.4375
  - o Is the treatment ongoing? = Yes
    - Has there been intensification? = Yes
      - (date of the first intensification index date)/30.4375
      - Has there been intensification? = No
        - Censured time: (date of the last assessment index date)/30.4375
- Perianal disease at diagnosis:
  - Fistulas at diagnosis=Yes and type=anal or rectovaginal -> Yes
  - Disease behaviour = Anal (CD patients) -> Yes
  - Other case -> No
- Previous abdominal surgeries:




Date: 17FEB2022

- Yes if Health resource utilization includes:
  - Any resection
  - Any resection with ostomy
  - Any resection with reservoir
  - Any stricturoplasty
- Reason end of first line:
- Wand Subject to the Applicable Terms of Use o Primary failure: "PNR: Without primary response"
  - Secondary failure: "SLR: Lost of response"
  - o Safety: "AE: Adverse Event"
  - Other:
    - "PR: Partial response"
    - "Remission"
    - "Other"
  - o Missing: "Unknown"

#### 7.2 Hypothesis and statistical methods

### 7.2.1 Univariate analysis. Descriptive statistics

Descriptive analysis of the collected variables will be carried out. Depending on the variable nature will be presented:

- Categorical variables will be summarized by frequencies and percentages.
- · Continuous variables will be summarized by means of central tendency and dispersion measures: mean, standard deviation, median, 25% and 75% (Q1 and Q3) percentiles and extreme values (minimum and maximum).

### 7.2.2 Bivariate analysis

When it is of interest to answer the study objectives, the relationship between variables will be evaluated:

- For two categorical variables, contingency tables with the frequency in each category and the percentage by columns will be presented. To evaluate the possible association Chi-square tests or Fisher's exact test will be performed and the resulting p-value will be presented.
- For a numerical variable with a categorical, descriptive statistics will be presented by groups. To evaluate the possible association, T-Test, ANOVA or Wilcoxon or Kruskal-Wallis nonparametric tests will be performed, as well as their resulting p-value.



| Study: EVOLVE |
|------------------|
| Date : 17FEB2022 |

To evaluate the relationship between two numerical variables, the Pearson or Spearman correlation will be presented, as well as its resulting p-value.

The methods described in section

The me

Only and Subject to the

- - o Other:
    - First line / Second line
- UC patients:
  - VDZ/Other
  - o VDZ:
    - First line / Second line
  - o Other:
    - First line / Second line

### 7.4.2 Endpoint analysis

Propensity scores inverse probability treatment weighting (PS-IPTW) will be used to ensure comparability between treatment groups (VDZ vs. Other biologic). 5 propensity scores will be estimated:

- CD patients
- UC patients
- CD with 1st line treatment
- UC with 1st line treatment
- CD with 2<sup>nd</sup> line treatment
- UC with 2<sup>nd</sup> line treatment

A logistic regression with treatment group as a response will be adjusted to estimate PS-IPTW, the model will include:

Age at index date (years)



| Study: EVOLVE |
|------------------|
| Date : 17FEB2022 |

Sex

- Disease duration (time between first ever CD/UC diagnosis and index data (years)) Aicable Terms of Use
- Smoking status at index date
- HBI score / Mayo score
- Perianal disease at diagnosis or index date (only CD patients)
- Previous abdominal surgeries
- Previous perianal surgeries
- Disease location
- Disease behaviour (only CD patients)
- Biologic treatment line (only with PS-IPTW for CD and UC patients)
- Any Corticosteroids treatment administered within the 6 months prior the index date
- Any Immunomodulators treatment administered within the 6 months prior the index date
- Logarithm of PCR (mg/L)
- Logarithm of Fecal calprotectin (mg/Kg)
- The patient has had extra intestinal manifestation within the 6 months prior the index
- Reason for discontinuation 1st line treatment (only for CD/UC 2nd line treatment patients)
  - Reasons for discontinuation will be pooled in the following way:
    - Primary failure
    - Secondary failure
    - Safety

The missing data of all variables will be imputed by using a multiple imputation method, see section 6.5.

A description of the variables without and with each PS-IPTW will be presented. A graphic with standardized means after and before each PS-IPTW (Love plot) will be presented. A density plot will be presented afet and before each PS-IPTW.

The distribution of each of the quantitative covariates included in the model after each PS-IPTW will be represented with boxplots.

#### List of endpoints:

Discontinuation. Percentage of patients with discontinuation. Logistic regression will be used.



| Study : EVOLVE |
|------------------|
| Date : 17FEB2022 |

Time to discontinuation. Median, p25 and p75 of time to discontinuation. Kaplan Meier and Log-Rank test will be used.

- Duration of treatment. Median, p25 and p75 of duration of treatment. Kaplan Meier and Log-Rank test will be used.
- Intensification. Percentage of patients with one or more intensification. Logistic regression will be used.
- Time to intensification. Median, p25 and p75 of time to discontinuation. Kaplan Meier and Log-Rank test will be used.
- Clinical response. Percentage of patients with clinical response. It will be evaluated at 14/52 weeks after index date. Logistic regression will be used.
- Clinical remission. Percentage of patients with clinical remission. It will be evaluated at 14/52 weeks after index date. Logistic regression will be used.
- Endoscopic response at 52 weeks. Percentage of patients with clinical response. Logistic regression will be used.
- Endoscopic remission at 52 weeks. Percentage of patients with clinical remission. Logistic regression will be used.
- Biochemical remission based on CPR. Percentage of patients with clinical remission. It will be evaluated at 14/52 weeks after index date. Logistic regression will be used.
- Biochemical remission based on fecal calcoprotein. Percentage of patients with clinical remission. It will be evaluated at 14/52 weeks after index date. Logistic regression will be used.

#### Each endpoint will be compare between:

- CD patients
  - VDZ 1st line Vs. VDZ 2nd line<sup>1</sup>
  - VDZ Ileal Vs. VDZ Colonic/Ileocolonic<sup>1</sup>
  - VDZ Ileal 1st line Vs. VDZ Colonic/Ileocolonic 1st line<sup>1</sup>
  - VDZ Ileal 2nd line Vs. VDZ Colonic/Ileocolonic 2nd line1
  - VDZ Ileal Intensification Vs. VDZ Colonic/Ileocolonic Intesification<sup>1</sup>
  - VDZ Ileal No Intensification Vs. VDZ Colonic/Ileocolonic No Intesification<sup>1</sup>
  - VDZ 2 years or more diagnosis Vs. VDZ less than 2 years diagnosis<sup>1</sup>
  - VDZ 2 years or more diagnosis 1st line Vs. VDZ less than 2 years diagnosis – 1st line¹
  - VDZ 2 years or more diagnosis 2nd line Vs. VDZ less than 2 years diagnosis – 2nd line¹
  - VDZ Inflamatory Vs. VDZ Stricturing/Penetrating<sup>1</sup>
  - VDZ Inflamatory 1st line Vs. VDZ Stricturing/Penetrating 1st line<sup>1</sup>



Study : EVOLVE Version : 6.0

Date: 17FEB2022

- o VDZ Inflamatory 2nd line Vs. VDZ Stricturing/Penetrating 2nd line1
- O.B. − 1st line Vs. O.B. − 2nd line¹
- o O.B. Ileal Vs. O.B. Colonic/Ileocolonic1
- O.B. Ileal 1st line Vs. O.B. Colonic/Ileocolonic 1st line<sup>1</sup>
- o O.B. Ileal 2nd line Vs. O.B. Colonic/Ileocolonic 2nd line1
- o O.B. Ileal Intensification Vs. O.B. Colonic/Ileocolonic Intesification1
- o O.B. Ileal No Intensification Vs. O.B. Colonic/Ileocolonic No Intesification<sup>1</sup>
- o O.B. 2 years or more diagnosis Vs. O.B. less than 2 years diagnosis
- O.B. − 2 years or more diagnosis − 1st line Vs. O.B. − less than 2 years diagnosis 1st line¹
- O.B. − 2 years or more diagnosis − 2nd line Vs. O.B. ► less than 2 years diagnosis 2nd line¹
- O.B. Inflamatory Vs. O.B. Stricturing/Penetrating<sup>1</sup>
- o O.B. Inflamatory 1st line Vs. O.B. Stricturing/Penetrating 1st line1
- o O.B. Inflamatory 2nd line Vs. O.B. Stricturing/Penetrating 2nd line1
- o VDZ Vs. O.B.<sup>2</sup>
- VDZ 1st line Vs. O.B. 1st line<sup>3</sup>
- o VDZ 2nd line Vs. O.B. 2nd line4
- o VDZ Colonic/Ileocolonic Vs. O.B. Colonic/Ileocolonic<sup>2</sup>
- o VDZ Colonic/Ileocolonic 1st line Vs. O.B. Colonic/Ileocolonic 1st line<sup>3</sup>
- ∨DZ Colonic/Ileocolonic 2nd line Vs. O.B. Colonic/Ileocolonic 2nd line<sup>4</sup>
- VDZ Ileal Vs. O.B. Ileal<sup>2</sup>
- ∨DZ Ileal 1st line Vs. O.B. Ileal 1st line³
- VDZ Ileal 2nd line Vs. O.B. Ileal 2nd line<sup>4</sup>
- VDZ less than 2 years diagnosis Vs. O.B. less than 2 years diagnosis²
- VDZ less than 2 years diagnosis 1st line Vs. O.B. less than 2 years diagnosis 1st line<sup>3</sup>
- $_{\odot}\,$  VDZ less than 2 years diagnosis 2nd line Vs. O.B. less than 2 years diagnosis 2nd line  $^{4}\,$
- VDZ 2 years or more diagnosis Vs. O.B. 2 years or more diagnosis<sup>2</sup>
- VDZ 2 years or more diagnosis 1st line Vs. O.B. 2 years or more diagnosis – 1st line<sup>3</sup>
- VDZ 2 years or more diagnosis 2nd line Vs. O.B. 2 years or more diagnosis – 2nd line<sup>4</sup>
- o VDZ Inflamatory Vs. O.B. Inflamatory <sup>2</sup>
- VDZ Inflamatory 1st line Vs. O.B. Inflamatory 1st line <sup>3</sup>



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

- VDZ Inflamatory 2nd line Vs. O.B. Inflamatory 2nd line <sup>4</sup>
- VDZ Stricturing/Penetrating Vs. O.B. Stricturing/Penetrating<sup>2</sup>
- o VDZ Stricturing/Penetrating 1st line Vs. O.B. Stricturing/Penetrating 1st line 3
- cable Terms of Use o VDZ Stricturing/Penetrating - 2nd line Vs. O.B. - Stricturing/Penetrating - 2nd line 4

#### UC

- VDZ 1st line Vs. VDZ 2nd line¹
- VDZ Extensive colitis Vs. VDZ Proctitis/Left colitis<sup>1</sup>
- VDZ Extensive colitis 1st line Vs. VDZ Proctitis/Left colitis 1st line<sup>1</sup>
- VDZ Extensive colitis 2nd line Vs. VDZ Proctitis/Left colitis 2nd line<sup>1</sup>
- o VDZ Extensive colitis Intensification Vs. VDZ Proctitis/Left colitis -Intesification1
- VDZ Extensive colitis No Intensification Vs. VDZ Proctitis/Left colitis No Intesification1
- VDZ 2 years or more diagnosis Vs. VDZ less than 2 years diagnosis<sup>1</sup>
- diagnosis - 1st line1
- VDZ 2 years or more diagnosis 2nd line Vs. VDZ less than 2 years diagnosis – 2nd line1
- O.B. − 1st line Vs. O.B. 2nd line¹
- O.B. Extensive colitis Vs. O.B. Proctitis/Left colitis<sup>1</sup>
- o O.B. Extensive colitis 1st line Vs. O.B. Proctitis/Left colitis 1st line1
- O.B. Extensive colitis 2nd line Vs. O.B. Proctitis/Left colitis 2nd line<sup>1</sup>
- o O.B. Extensive colitis Intensification Vs. O.B. Proctitis/Left colitis -Intesification<sup>1</sup>
- O.B. Extensive colitis No Intensification Vs. O.B. Proctitis/Left colitis No Intesification1
- O.B. 2 years or more diagnosis Vs. O.B. less than 2 years diagnosis<sup>1</sup>
- O.B. 2 years or more diagnosis 1st line Vs. O.B. less than 2 years diagnosis 1st line1
- o O.B. 2 years or more diagnosis 2nd line Vs. O.B. less than 2 years diagnosis 2nd line1
- o VDZ Vs. O.B.5
- VDZ 1st line Vs. O.B. 1st line<sup>6</sup>
- VDZ 2nd line Vs. O.B. 2nd line<sup>7</sup>
- VDZ Proctitis/Left colitis Vs. O.B. Proctitis/Left colitis<sup>5</sup>



Study : EVOLVE


Date: 17FEB2022

- o VDZ Proctitis/Left colitis 1st line Vs. O.B. Proctitis/Left colitis 1st line<sup>6</sup>
- o VDZ Proctitis/Left colitis 2nd line Vs. O.B. Proctitis/Left colitis 2nd line<sup>7</sup>
- VDZ Extensive colitis Vs. O.B. Extensive colitis<sup>5</sup>
- VDZ Extensive colitis 1st line Vs. O.B. Extensive colitis 1st line<sup>6</sup>
- ∨DZ Extensive colitis 2nd line Vs. O.B. Extensive colitis 2nd line<sup>7</sup>
- ∨DZ less than 2 years diagnosis Vs. O.B. less than 2 years diagnosis<sup>5</sup>
- VDZ less than 2 years diagnosis 1st line Vs. O.B. less than 2 years diagnosis – 1st line<sup>6</sup>
- VDZ less than 2 years diagnosis 2nd line Vs. O.B. less than 2 years diagnosis – 2nd line<sup>7</sup>
- VDZ 2 years or more diagnosis Vs. O.B. 2 years or more diagnosis<sup>5</sup>
- VDZ 2 years or more diagnosis 1st line Vs. O.B. 2 years or more diagnosis 1st line<sup>6</sup>
- VDZ 2 years or more diagnosis 2nd line Vs. O.B. 2 years or more diagnosis - 2nd line<sup>7</sup>
- ¹Data without PS-IPTW.
- <sup>2</sup>Data with PS-IPTW (CD).
- <sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).
- <sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).
- 5Data with PS-IPTW (UC).
- <sup>6</sup>Data with PS-IPTW (UC-1st line)
- <sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

Per each endpoint a table with all the comparisons will be presented. The table will contain:

- Endpoint of each group of the comparison.
- Number of patients analysed per group of the comparison
- OR (only percentage endpoints)
- P-value.

For each time to event comparison a figure with Kaplan-Meier's curves will presented.

Also a multivariate logistic regression will be performed for Discontinuation, One intensification or more, clinical response at 52 weeks and clinical remission at 52 weeks. The logistic regression will be performed separated by treatment group (VDZ and Other Biologic patients) and disease (CD and UC patients). Exploratory variables:

- Line of treatment
- Disease location
- Time between first ever CD/UC diagnosis and index date



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

- Disease behaviour (only CD patients)
- All interactions

The PROC MIANALYSE (SAS software 9.4 or posterior) will be used in all analyses.

### 7.5 Analysis of secondary objectives

- Characterize patients treated with VDZ or other biologics (infliximab, adalimumab, or golimumab [UC only]) as first and second line biologic therapy in terms of demographics, medical, and treatment histories.

View section 7.3.

- Describe the real world clinical effectiveness of VDZ vs. other biologics at least 12 months post-treatment initiation (in a subgroup of patients with adequate follow-up available).

Included in section 7.4.

- Describe the safety events occurring post biologic treatment initiation (VDZ or other biologics).

The incidence (%) and rate incidence (per 100 patient-year) of adverse events, serious adverse events, related with index treatment adverse events and related with index treatment serious adverse events, infections, serious infections and malignancies will be presented per each disease group (UC/DC).

The incidence and rate incidence will be compared between:

- CD patients
  - VDZ Vs. Other Biologic<sup>1</sup>
  - VDZ 1st line Vs. Other Biologic 1st line<sup>1</sup>
  - o VDZ 2nd line Vs. Other Biologic 2nd line<sup>2</sup>
- UC patients
  - VDZ Vs. Other Biologic<sup>3</sup>
  - VDZ 1st line Vs. Other Biologic 1st line<sup>3</sup>
  - $\circ$  VDZ 2nd line Vs. Other Biologic 2nd line<sup>4</sup>

Data with PS-IPTW (CD)

<sup>2</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line)

<sup>3</sup>Data with PS-IPTW (UC)

<sup>4</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line)

The incidence comparisons will be estimated by using a logistic regression.

The incidence rate comparisons will be estimated by using a Poisson regression.

Per each AA type and incidence/incidence rate a table with all the comparisons will be presented. The table will contain:



| Study: EVOLVE |
|------------------|
| Date : 17FEB2022 |

Incidence/Incidence rate of each group of the comparison.

- OR (incidence) or RR (incidence rate)
- P-value.

o Number and percentage of patients with an AF

- Number of adverse events.
- Numbers of adverse events by:
  - Seriousness (Resulted in death / Was life-threatening / Required in patient hospitalization or prolongation of existing hospitalization / Resulted in persistent or significant disability or incapacity / Was a congenital anomaly or birth defect / Was an important medical event / None of the above)
  - Related to index drug (Yes / No)
  - Event Resolved (Yes (Duration) / No / Unknown)
  - Action taken with index drug (Treatment withdrawn / Dose reduced / Dose increased / Dose delayed / Dose not changed / Unknown / Not applicable)
  - Outcome (Recovered / Not recovered / Fatal / Recovering / Recovered with sequelae (Unknown)
  - Duration (days)

The PROC MIANALYSE (SAS software 9.4 or posterior) will be used in all analyses with PS-IPTW data.

Quantify healthcare resource utilization including the rates of healthcare professional (HCP) and emergency department (ED) visits, hospitalizations and Inflammatory Bowel Disease (IBD) related surgical procedures.

Descriptive analysis of visits during the 12 months prior index date (index date included) and 12 months post-index date will be performed.





 ${\bf Study:EVOLVE}$ Version: 6.0

Date: 17FEB2022





### 9. Results

### 9.1 Study population

Table 1.1.1 Patients recruited, valid and excluded

| | | | | 70 |
|---|---|---|---|---|
| | | | | Patients |
| | | Total | Patients | recruited |
| | | patients | recruited | with Other |
| | | recruited | with VDZ | Biologic |
| | | (n=xx) | (n=xx) | (n=xx) |
| Valid patients | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Excluded patients | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ( | Silly, | | |
| Reason of exclusion*: | and | | | |
| Patients without a diagnosis of moderate to severe UC or | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| CD documented in the medical chart | | | | |
| Patients that have not received any dose of VDZ or other | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| biologic (infliximab, adalimumab, or golimumab [UC only]) | | | | |
| during the eligibility period | | | | |
| Patients younger than 18 years of age at the time of | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| treatment initiation with VDZ or other biologic (index event) | | | | |
| Patients that have not received the biologic treatment as | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| first-line or second-line treatment for UC or CD | | | | |
| Patients without a minimum of six months of follow up | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| between index date and date of chart abstraction initiation | ( ) | , | , | , |
| | (0/) | ( | ( 0( ) | ( 0( ) |
| Patients that received VDZ or another biologic as part of an | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| interventional clinical trial ever in their lifetime (includes index | | | | |
| (treatment) | | | | |
| Patients that initiated index treatment as combination | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| therapy with two biologic agents | | | | |
| Patients that the biologic was prescribed for the treatment | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| of perianal disease | | | | |
| Patients that have received a biologic prior to the index | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| period for a disease other than inflammatory bowel disease | | | | |



| Study: EVOLVE |
|------------------|
| Date : 17FEB2022 |

**Patients** recruited **Patients Total** recruited patients with VDZ recruited (n=xx) (n=xx) Patients with clinical record unavailable n (%) xx ( xx.x%) xx ( xx.x%)

#### Table 1.1.2 Follow-up

| | 1 4510 11 | rabio ii ii z i olioti ap | | |
|---|---|---|---|---|
| | | Total patients | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) | (n=xx) |
| Time of follow-up (months) | n | xx | XX | XX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Missing | OU XX | xx | xx |
| | .69 | 2 | | |
| Patients with at least 12 mo | nths | | | |
| of follow-up | , cio | | | |
| Total no-missing | nths | xx | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx | XX |
| Missing Missing | | | | |

<sup>\*</sup>The patients could present more than one reason.



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

### 9.2 Descriptive analysis

### 9.2.1 Groups description

Table 2.1.1 Groups and subgroups

| Table 2.1.1 Gloc | ips and subgroups | |
|---|---|---|
| | | Total |
| | | (n=xx) |
| Overall | | .:C3/0, |
| Treatment group | | POPIL |
| Total no-missing | n | xx |
| VDZ | n (%) | xx ( xx.x%) |
| Other biologic | n (%) | xx ( xx.x%) |
| Missing | n SUP, | xx |
| Disease | and | |
| Total no-missing | KA | xx |
| CD © | n (%) | xx ( xx.x%) |
| UC | n (%) | xx ( xx.x%) |
| Missing | n | xx |
| Treatment line | | |
| Total no-missing | n | xx |
| 1 <sup>st</sup> 40 <sup>f</sup> f | n (%) | xx ( xx.x%) |
| 2 <sup>nd</sup> | n (%) | xx ( xx.x%) |
| Missing | n | xx |
| Overall Treatment group Total no-missing VDZ Other biologic Missing Disease Total no-missing CD UC Missing Treatment line Total no-missing 1st 2nd Missing WDV Disease Total no-missing | | |
| Disease | | |
| Total no-missing | n | XX |
| CD | n (%) | xx ( xx.x%) |
| UC | n (%) | xx ( xx.x%) |
| Missing | n | xx |


Study : EVOLVE


Date : 17FEB2022

n n(%) n (%) n (%) and subject to the population of the population Treatment line Total no-missing 1<sup>st</sup>  $2^{nd}$ Missing Other biologic Disease Total no-missing CD UC Missing Treatment line Total no-missing 1<sup>st</sup> 2<sup>nd</sup> Missing CD Treatment group Other biologic
Missing n XXn (%) xx ( xx.x%) n (%) xx ( xx.x%) n XX Total no-missing n ХX 1<sup>st</sup> n (%) xx ( xx.x%)



 $2^{\text{nd}}$ 

### STATISTICAL ANALYSIS PLAN

Study : EVOLVE


Date : 17FEB2022

n and Subject to the Reputable Territor of Use of the Reputable Territor of Use of the Reputable Territor of the Reputable Total Treatment line Total no-missing n XX1<sup>st</sup> n (%) xx ( xx.x%)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

n (%)

xx ( xx.x%)



Study : EVOLVE


Date : 17FEB2022

| Missing | n | xx |
|---|---|---|
| imoonig | " | <b>,</b> ,, |
| UC-VDZ | | xx |
| Treatment line | | è, |
| Total no-missing | n | xx apple |
| 1 <sup>st</sup> | n (%) | xx (xx.x%) |
| 2 <sup>nd</sup> | n (%) | xx ( xx.x%) |
| Missing | n | xx xx |
| UQ Qdhaa bialaata | n (%) n (%) n n | ŞÖ. |
| UC-Other biologic Treatment line | 3501 | |
| | | xx |
| 1 otal 110-11116581119 | On (%) | xx ( xx.x%) |
| 2 <sup>nd</sup> | n (%) | xx ( xx.x%) |
| Missing | n | xx |
| Total no-missing 1st 2nd Missing | | |



Study: EVOLVE STATISTICAL ANALYSIS PLAN Version: 6.0

Date: 17FEB2022

# 9.2.2 By treatment

| | Table 2.2.1 Demogra | ble 2.2.1 Demographics | |
|---|---|---|---|
| | | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) |
| Sex | | | (8) |
| Total no-missing | n | XX | i Calo |
| Male | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx 10 | xx |
| Age at index date (years) | n | sulipecitio s | xx |
| | Mean (SD) | XX.X (XX.X) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | XX | xx |
| | CO. | | |
| BMI (Kg/m²) | W <sub>©</sub> , u | xx | xx |
| COL | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| John | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| 1.01 | Min, Max | xx, xx | xx, xx |
| BMI (Kg/m²) Smoking status at index treatment initial | Missing | xx | xx |
| Smoking status at index treatment initi | iation | | |
| Total no-missing | n | XX | xx |
| Never smoked | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Former smoker | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Current smoker | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | XX | xx |



Study : EVOLVE


Date : 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Number of years that the patient has smoked <sup>1</sup> | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | xx | bb xx |
| | | "IN | S |
| Number of years that the patient has been smoked <sup>2</sup> | n | xx.x (xx.x, xx.x) xx, xx | xx |
| | Mean (SD) | Cxx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x)<br>xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | xx | xx |
| Cigarettes per day² Work status at index date | n | xx | xx |
| affilh | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| COV | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| 4011 | Min, Max | XX, XX | xx, xx |
| 60( ) | Missing | XX | XX |
| Work status at index date | | | |
| Total no-missing | n | xx | xx |
| Unemployed | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Retired | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Home maker | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Full-time employee | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | , , | |



Study : EVOLVE


Date : 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Full-time student | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Part-time student | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Disability/sick leave | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| Number of days the patient has been on sick leave within the 6 months prior to the index date | n | xx | Applicable |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | S <sup>U</sup> xx, xx | xx, xx |
| | Missing | xx xx | xx |

<sup>&</sup>lt;sup>1</sup> Former smoker patients.

Table 2.2.2 Disease Characteristics - CD patients

| amerc | | VDZ | Other Biologic |
|---|---|---|---|
| Mill | | (n=xx) | (n=xx) |
| Age at first ever CD diagnosis (years) | n | XX | xx |
| 401, | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Kok | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| da. | Min, Max | xx, xx | xx, xx |
| Age at first ever CD diagnosis (years) | Missing | xx | XX |
| Location of intestinal involvement at diagnosis* | | | |
| Total no-missing | n | xx | xx |
| lleal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Colonic | n (%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>2</sup> Current smoker patients.



Study : EVOLVE


Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Upper GI tract | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| lleocolonic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | XX | xx xx xx |
| Type of disease behaviour at diagnosis | 5* | | is able |
| Total no-missing | n | xx | Obli xx |
| Inflammatory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Stricturing | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Penetrating | n (%) | xx ( xx.x%) xx ( xx.x%) xx xx xx ( xx.x%) | xx ( xx.x%) |
| Anal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| Active fistulas at diagnosis | O// | | |
| Total no-missing | n 150 | xx | xx |
| Yes | (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Total no-missing Yes No Missing Type of active fistulas at diagnosis*1 | n | XX | xx |
| Γype of active fistulas at diagnosis* <sup>1</sup> | | | |
| Total no-missing | n | xx | xx |
| Anal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Rectovaginal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Enterocutaneous | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Internal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| Number of fistulas | | | |



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

| | VDZ | Other Biologic |
|-----------------|-------------------|-------------------|
| | (n=xx) | (n=xx) |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Min, Max | xx, xx | xx, xx |
| Missing | xx | xx < |

<sup>&</sup>lt;sup>1</sup> Patients with active fistulas.

Table 2.2.3 Disease Activity - CD patients

| | 2.00000710117119 | or patients | |
|---|---|---|---|
| | | VDZ VO | Other Biologic |
| | | (n=xx) | (n=xx) |
| Time between index date and assessment (months) | n | Supx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| Ċ | Missing | xx | xx |
| HBI score registered in the medical chart? Total no-missing | n | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Total no-missing Yes No Missing | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | XX | xx |
| Can any subscale of HBI be extracted from medical chart? <sup>1</sup> | | | |
| Total no-missing | n | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | XX |

<sup>\*</sup> More than an answer possible.



Study : EVOLVE


Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| eneral well being <sup>2</sup> | | | xx<br>xx ( xx.x%) |
| Total no-missing | n | xx | xx |
| Unknown | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Vell or very well | n (%) | xx ( xx.x%) | xx ( xx x%) |
| Slightly below par | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Poor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| /ery poor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Terrible | n (%) | xx ( xx.x%) xx ( xx.x%) xx xx | xx ( xx.x%) |
| Missing | n | C/I/Oxx | xx |
| | < | 40 | |
| odominal pain <sup>2</sup> | 143 | | |
| Total no-missing | n Offi | xx | xx |
| lone | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1ild | (%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None Mild Moderate Severe Missing | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| ımber of liquid or soft stools per day² | n | xx | xx |
| 169,0 | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| < 3L | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| umber of liquid or soft stools per day <sup>2</sup> | Min, Max | XX, XX | xx, xx |
| | Missing | xx | xx |
| bdominal mass <sup>2</sup> | | | |
| otal no-missing | n | xx | xx |



Study : EVOLVE

Date: 17FEB2022


| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| None | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Questionable or dubious definite | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Definite and tender | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx . C |
| | | | able |
| Complications <sup>2*</sup> | | | xx |
| Total no-missing | n | xx | xx |
| None | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Erythema nodosum | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Pyoderma gangrenosum | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other bowel-related fistula | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| New fistula | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Arthritis or arthralgia | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Apthous ulcers | n.(%) | xx ( xx.x%) | xx ( xx.x%) |
| Anal fissure, fistula or perirectal abscess | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Febrile (fever) episode over 100 degrees | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| during past week | | | |
| Abscess | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Iritis or uveitis | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| 98. | | | |
| Abscess Iritis or uveitis Missing HBI overall score <sup>3</sup> | n | xx | xx |
| of the second se | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | XX | xx |
| SES-CD score | n | xx | xx |




Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | xx | XX.X (XX.X, XX.X) XX, XX XX XX XX XX XX |
| | | | aldie |
| Patient status according to physician | | | OPILO |
| assessment | | | Dr. |
| Total no-missing | n | xx ill | xx |
| Remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Partial remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Not in remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n ? | xx | xx |

<sup>\*</sup> More than an answer possible.

<sup>&</sup>lt;sup>1</sup> Patients without HBI score registered in the medical chart.

Jistered Jistered Aredai. For Non-Commer Property of Fakedai. <sup>2</sup> Patients with subscales of HBI registered in medical chart.

<sup>&</sup>lt;sup>3</sup> Patients with HBI score registered or calculated.




Date: 17FEB2022

Table 2.2.4 Disease Characteristics – UC patients

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Age at first ever UC diagnosis (years) | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xxı xx |
| | Missing | xx | POS xx |
| | | 110 | <b>3</b> ' |
| Location of UC at diagnosis* | | 40 | |
| Total no-missing | n | xx, xx xx | xx |
| Proctitis/proctosigmoiditis | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Left-sided (distal to splenic flexure) | n (%)<br>n (%)<br>n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Extensive colitis (proximal to hepatic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| flexure) | 01 | | |
| Unspecified | n(%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

Table 2.2.5 Disease Activity – UC patients

| 20,00 | | VDZ | Other Biologic |
|---|---|---|---|
| 40, | | (n=xx) | (n=xx) |
| Time between index date and assessment | n | XX | xx |
| (months) | | | |
| it akeor | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX | xx, xx |
| | Missing | xx | xx |

Partial Mayo score registered in the medical chart?



Study : EVOLVE

Date: 17FEB2022


| | | VDZ | Other Biologic |
|---|---|---|---|
| Total na mainain n | | (n=xx) | (n=xx) |
| Total no-missing | n | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| | | | 6301 |
| Can any subscore of PMS be extracted from | | | adilo |
| medical chart?1 | | | DO, |
| Total no-missing | n | xx H | xx (xx.x%) xx xx xx xx |
| Yes | n (%) | XX ( XX.X70) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx xx | xx |
| | , of | | |
| Stool frequency <sup>2</sup> | n (%) n n (%) | | |
| Total no-missing | n S | XX | XX |
| Unknown | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Normal number of stools for subject | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1-2 stools per day more than normal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 3-4 stools per day more than normal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| >=5 stools per day more than normal | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| 9.9. | | | |
| Rectal bleeding <sup>2</sup> | | | |
| Total no-missing | n | xx | xx |
| No blood seen | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Streaks of blood with stool less than half the | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| time | | | |
| Obvious blood with stool most of the time | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Blood alone passes | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE


Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Missing | n | xx | xx |
| Physician global assessment <sup>2</sup> | | | |
| Total no-missing | n | xx | xx Cl |
| Normal or remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild disease | n (%) | xx ( xx.x%) | × ( xx.x%) |
| Moderate disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx (xx.x) | XX |
| | | Siloi | |
| Partial Mayo overall score <sup>3</sup> | n | xx b | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| 4 | Missing | xx | xx |
| alle | | | |
| Patient status according to physicia | ın | | |
| assessment | | | |
| Total no-missing | n | xx | xx |
| Remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Partial remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Not/in remission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

- \* More than an answer possible.
  - <sup>1</sup> Patients without partial Mayo score registered in the medical chart.
  - <sup>2</sup> Patients with subscores of PMS registered in medical chart.
  - <sup>3</sup> Patients with partial Mayo score registered or calculated.




Date: 17FEB2022

# Table 2.2.6 Diagnostic imaging

| | VDZ | Other Biologic |
|-------|-------------------------------------|--------------------------|
| | | Guioi Biologio |
| | (n=xx) | (n=xx) |
| n | xx | Other Biologic<br>(n=xx) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx (xx.x%) |
| n | xx | Poly, xx |
| | *** | 2 |
| | *** | |
| n | iw Ce | xx |
| n (%) | | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n 😞 | xx | xx |
| 1/23 | | |
| , Co | | |
| | n (%) n (%) n n n n (%) n (%) n (%) | n (%) |



Study : EVOLVE

Date: 17FEB2022


Table 2.2.7 Laboratory determinations



Study : EVOLVE

Date: 17FEB2022


# **Table 2.2.8 Extra Intestinal Manifestations**

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| The patient has had extra inte manifestation within the 6 months pricindex date? | stinal<br>or the | | |
| Total no-missing | n | xx | ×XOIE |
| Yes | n (%) | xx ( xx.x%) | xxx ( xxx x0/. ) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx (xx.x%) xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx (xx.x%) | xx |
| Disease*1 | | Subject | |
| Total no-missing | n | xx | xx |
| Axial arthropathy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Peripheral arthropathy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Erythema nodosum | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Pyoderma gangrenosum | (%) | xx ( xx.x%) | xx ( xx.x%) |
| Sweet's syndrome | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Pyoderma gangrenosum Sweet's syndrome Oral alphthous ulcers Episcleritis Uveitis PSC | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Episcleritis | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Uveitis | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| PSC | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| o <sup>X</sup> | | | |
| Intensity*2 | | | |
| Total no-missing | n | xx | xx |
| Mild | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | n (%) | xx ( xx.x%) | xx ( xx.x%) |



| Study : EVOLVE |
|------------------|
| Date : 17FEB2022 |

| Missing n xx xx Ongoing at index date?² Total no-missing n xx xx xx Yes n (%) xx (xxx%) xx (xxx%) No n (%) xx (xxx%) xx (xxx%) Missing n xx xx xx 1Patients with extra intestinal manifestation. *Almost one extra intestinal manifestation. * More than an answer possible. | | | VDZ<br>(n=xx) | Other Biologic<br>(n=xx) |
|---|---|---|---|---|
| Yes n (%) xx ( xx.x%) xx ( xx.x%) | Missing | n | | |
| Yes n (%) xx ( xx.x%) xx ( xx.x%) | Ongoing at index date? <sup>2</sup> | | | |
| Yes n (%) xx ( xx.x%) xx ( xx.x%) | Total no-missing | n | xx | xx . C |
| Missing n xx 1Patients with extra intestinal manifestation. 2Almost one extra intestinal manifestation. * More than an answer possible. Only and Subject to the possible of the possible of the possible of the possible on the possible on the possible on the possible on the possible of the possible of the possible on the possible of the possible | Yes | n (%) | xx ( xx.x%) | 101 |
| 1Patients with extra intestinal manifestation. 2Almost one extra intestinal manifestation. * More than an answer possible. | No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1Patients with extra intestinal manifestation. 2Almost one extra intestinal manifestation. * More than an answer possible. Only and Subject to the commercial use only and Subject to the commercial use of the commercial | Missing | n | xx | XX XX |
| <sup>2</sup> Almost one extra intestinal manifestation. * More than an answer possible. * More than an answer possible. Only and Subject the O | <sup>1</sup> Patients with extra intestir | nal manifestation. | 11/2 | 9 |
| * More than an answer possible. *More than an an answer possible. *More than an an answer possible. *More than an an answer possible. *More than an a | <sup>2</sup> Almost one extra intestina | al manifestation. | -Ci | |
| atty of Takeda. For | 40n.c | Ohmercia | | |
| | co's | | | |
| | attl of takeda. | | | |



Study : EVOLVE

Date : 17FEB2022


# Table 2.2.9 Comorbid medical conditions

| Table 2.2 | .9 Comorbia | medical conditions | |
|---|---|---|---|
| | | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) |
| The patient has had comorbid medical condition within the 6 months prior the independent date? | | | ×ole (ex |
| Total no-missing | n | xx | ×O/E |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx iii | xx |
| Disease*1 | | xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx (xx.x%) | |
| Total no-missing | n | xx | xx |
| Myocardial infection | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| CHF | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Peripheral vascular disease | n (%)5 | xx ( xx.x%) | xx ( xx.x%) |
| CVA or TIA | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dementia | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| CVA or TIA Dementia CPPD Connective tissue disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Connective tissue disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Peptic ulcer disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Liver disease | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Diabetes mellitus | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hemiplegia | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate to severe CKD | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Solid tumor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Leukemia | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Lymphoma | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| AIDS | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |




Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | |
| Missing | n | XX | xx |
| Intensity* <sup>2</sup> | | | (n=xx) |
| Total no-missing | n | xx | xx < |
| Mild | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx xo | xx |
| Ongoing at index date? <sup>2</sup> | | xx (xx.x%) xx xx (xx.x%) xx (xx.x%) | |
| Total no-missing | n | , d xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n S | xx | xx |
| <sup>1</sup> Patients with comorbid medic | al condition. | | |
| <sup>2</sup> Almost one comorbid medical | condition. | | |
| * More than an answer possible | e. | | |
| of Takeda. For Non.co. | | | |

<sup>&</sup>lt;sup>1</sup>Patients with comorbid medical condition.

<sup>&</sup>lt;sup>2</sup>Almost one comorbid medical condition.



Study : EVOLVE

Date: 17FEB2022


# Table 2.2.10Biologic treatment pre index treatment

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Fime between induction and index date months) | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |
| | Missing | xx *********************************** | xx |
| Fime between induction and maintenance weeks) | n | xx to the | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |
| | Missing | xx | xx |
| Has there been intensification? | | | |
| Has there been intensification? Total no-missing Yes | n | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| increase the dose. | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Decrease the frequency <sup>1</sup> | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Both <sup>1</sup> | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Decrease the frequency <sup>1</sup> Both <sup>1</sup> No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| ime between induction and intensification months) <sup>1</sup> | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |




Date: 17FEB2022

VDZ Other Biologic (n=xx)(n=xx)Missing хх XX

Time between induction and discontinuation (months)

| Mean (SD) | xx.x (xx.x) |
|-----------|-------------|

XX, XX

XX

xx ( xx.x%)

| Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
|-----------------|-------------------|-------------------|
| | | 4 1 1 |

XX

Missing XX

XX

### Reason for discontinuation

Total no-missing

| Without primary response | n (%) |
|--------------------------|-------|
| Lost of response | n (%) |

xx ( xx.x%)

| Partial response | n (%) | xx ( xx.x%) | xx ( xx.x%) |
|------------------|-------|-------------|-------------|
| Adverse event | n (%) | xx ( xx.x%) | xx ( xx.x%) |

Min, Max

n

Missing

1 Patients with intensification.

Property of Trakedai. xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) XX



Study : EVOLVE

Date: 17FEB2022


# Table 2.2.11Non-biologic treatment

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Any non-biologic treatment admini | stered | | |
| within the 6 months prior the index date | | | |
| Total no-missing | n | xx | xx |
| Yes | n (%) | xx ( xx.x%) | xx ( xx x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx ( xx.x%) xx ( xx.x%) xx xx ( xx.x%) xx xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | Ø xx |
| Type*1 | | iect | |
| Total no-missing | n | Silox | xx |
| Corticosteroids | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Immunomodulators | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Ant biotics | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – ASA | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 – ASA Other Missing Ongoing at index date? | n n | xx | xx |
| Coll | | | |
| Ongoing at index date?1 | | | |
| Total no-missing | n | xx | xx |
| Yes <sup>2</sup> | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No Leo | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

Patients with non-biologic treatment.

<sup>&</sup>lt;sup>2</sup>Almost one non-biologic treatment.

<sup>\*</sup> More than an answer possible.




Date: 17FEB2022

# Table 2.2.12End of study

| | | | VDZ | Other Biologic |
|---|---|---|---|---|
| | | | (n=xx) | (n=xx) |
| Has the patient prematurely | finished the stud | ly | | |
| Total no-missing | | n | xx | XX 🗷 |
| Yes | | n (%) | xx ( xx.x%) | xx (_xx.x%) |
| No | | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | | n | xx | S xx |
| Reason | | | xx (xx.x%) xx xx | |
| Total no-missing | | n | Silox | xx |
| Screening failure | | n (%) | xx (xx.x%) xx (xx.x%) | xx ( xx.x%) |
| AE | | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Patient decision | | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawn consent | | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Doctor's decision | <b>.</b> | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | ame | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | Cou. | n | XX | xx |
| Patient decision Withdrawn consent Doctor's decision Other Missing | 401 | | | |



| Study: EVOLVE |
|---------------|

Date: 17FEB2022

# 9.2.3 By treatment (CD patients)

# Table 2.3.1 Demographics (CD patients)

| | | VDZ | Other Biologic |
|------------------|-------|-------------|----------------|
| | | (n=xx) | (n=xx) |
| Sex | | | 40 |
| Total no-missing | n | xx | xx Ø |
| Male | n (%) | xx ( xx.x%) | xx (-xx.x%) |
| Female | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | ⊗ xx |
| | | .0 | |

Table 2.4.1 Demographics (CD-VDZ patients)

| 9.2.4 By treatment line (CD-VDZ patients) | | | |
|---|---|---|---|
| | \se | | |
| Table | 2.4.1 Demographics | (CD-VDZ patients) | |
| | Cio | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
| | we. | (n=xx) | (n=xx) |
| Sex | | | |
| Total no-missing Male | n | xx | xx |
| Male | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |



| S | tudy : EVOLVE |
|---|---------------|

Date: 17FEB2022

# 9.2.5 By treatment line (CD-Other Biologic Patients)

Table 2.5.1 Demographics (CD-Other Biologic patients)

| | | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
|------------------|-------------|----------------------|----------------------|
| | | (n=xx) | (n=xx) |
| ex | | | 10 |
| Total no-missing | n | xx | i Calo |
| Male | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx xo | XX |
| | | xx to the | |
| | | eno, | |
| | | 70 | |
| | | Jand S | |
| | C patients) | • | |

# 9.2.6 By treatment (UC patients)

Table 2.6.1 Demographics (UC patients)

| ue <sub>lo</sub> . | (n=xx) | (n=xx) |
|--------------------|----------------|-------------|
| n | xx | xx |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n | xx | xx |
| | n (%)<br>n (%) | n (%) |



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

# 9.2.7 By treatment line (UC-VDZ patients)

Table 2.7.1 Demographics (UC-VDZ patients)

| | | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
|------------------|-------|----------------------|----------------------|
| | | (n=xx) | (n=xx) |
| Sex | | | 10 |
| Total no-missing | n | xx | i Cal |
| Male | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx 10 | xx |
| | | biecit | |
| | | CIO | |

• • •

# 9.2.8 By treatment line (UC-Other Biologic Patients)

Table 2.8.1 Demographics (UC-Other Biologic patients)

| 0.1 | | |
|-------|----------------------|------------------------------------------|
| Mele | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
| | (n=xx) | (n=xx) |
| n | xx | XX |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n | xx | XX |
| | n<br>n (%)<br>n (%) | n xx n (%) xx ( xx.x%) n (%) xx ( xx.x%) |

...



Study : EVOLVE


Date: 17FEB2022

# 9.3 Primary Objective (Descriptive analysis)

# 9.3.1 Descriptive by treatment

Table 3.1.1 Biologic index treatment I

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | VDZ<br>(n=xx) | (n=xx) |
| Steroid status at index date | | (1. 7.2.) | 70/6 |
| Steroid Status at Index date | | | dico |
| Total no-missing | n | XX | PGK xx |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | alliq xx | xx |
| | 415 | 3 | |
| Main reason for starting biologic treatment at index | 0/, | | |
| date | 5 | | |
| Total no-missing | n | xx | xx |
| Lack of/incomplete UC or CD response to prior non- | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| biologic therapy | | | |
| Poor tolerability to prior non biologic therapy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of response to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Loss of response to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Partial response to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Poor tolerability to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Post-operative prophylaxis | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Subject choice | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Anticipated superior efficacy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Anticipated superior safety | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other Biologic contraindicated or not elig ble | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Route of administration | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE

Date : 17FEB2022


| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Confidence in using biologic without concomitant immunomodulator | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx \@{\ |
| | | | able |
| Reason for starting biologic treatment at index date * | | | dico |
| Total no-missing | n | xx | xx (xx.x%) |
| Lack of/incomplete UC or CD response to prior non- | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| biologic therapy | | -CL | |
| Poor tolerability to prior non biologic therapy | n (%) | xx ( xx x%) | xx ( xx.x%) |
| Lack of response to a prior Biologic | n (%) | C xx ( xx.x%) | xx ( xx.x%) |
| Loss of response to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Partial response to a prior Biologic | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Poor tolerability to a prior Biologic | on (%) | xx ( xx.x%) | xx ( xx.x%) |
| Poor tolerability to a prior Biologic Post-operative prophylaxis Subject choice Anticipated superior efficacy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Subject choice | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Anticipated superior efficacy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Anticipated superior safety | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Other Biologic contraindicated or not elig ble | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Route of administration | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Confidence in using biologic without concomitant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| immunomodulator | | | |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

<sup>\*</sup> More than an answer possible.



Study : EVOLVE

Date: 17FEB2022


Table 3.1.2 Biologic index treatment II

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Type of biologic | | | (n=xx) |
| Total no-missing | n | | xx |
| Original | n (%) | | xx ( xx.x%) |
| Infliximab | n (%) | | xx (xx.x%) |
| Biosimilar | n (%) | nd Suldiect to the | xx ( xx.x%) |
| Adalimumab | n (%) | Ni. | xx ( xx.x%) |
| Golimumab | n (%) | 2,40 | xx ( xx.x%) |
| Missing | n | Nie C | xx |
| | | SUL | |
| Posology (mg) (Induction) | n | xx | xx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | XX, XX | XX, XX |
| Q. | Missing | xx | xx |
| osology (mg) (Maintenance) | | | |
| osology (mg) (Maintenance) | n | xx | xx |
| 4011 | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Posology (mg) (Maintenance) | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| 80. | Min, Max | xx, xx | XX, XX |
| Kakeda. | Missing | xx | xx |
| ime between induction and maintenance | n | XX | XX |
| veeks) | | | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |



Study : EVOLVE


Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| | Missing | xx | xx |
| the treatment ongoing? | | | |
| Total no-missing | n | xx | XX C |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx ( xx.x%) xx ( xx.x%) xx xx ( xx.x%) |
| | | 70 | |
| eason for discontinuation <sup>2</sup> | | · ect | |
| Total no-missing | n | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx |
| Nithout primary response | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Loss of response | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Partial response | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Adverse event | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Remission | . (2) | xx ( xx.x%) | xx ( xx.x%) |
| Other | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Remission Other Missing | n | XX | xx |
| 400 | | | |
| as the patient take a new biologion at the patient and the patient are a second control of the patient and the patient are also becomes a second control of the patient are also becomes | С | | |
| Total no-missing | n | xx | xx |
| Yes X | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| me between index treatment and nev | v n | xx | XX |
| eatment (months) <sup>3</sup> | • " | ^^ | ^^ |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

xx.x (xx.x)

xx.x (xx.x)

Mean (SD)




Date: 17FEB2022

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | xx | xx Kelly |
| Posology (mg) (New treatment induction) <sup>3</sup> | n | xx | xx delle |
| | Mean (SD) | xx.x (xx.x) | ( , , , , , ) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | xx | xx |
| | | CIO | |
| Type of biologic <sup>3</sup> | ٠ | d | |
| Total no-missing | n N | xx.x (xx.x, xx.x) xx, xx | XX |
| VDZ | n (%) | | xx ( xx.x%) |
| Infliximab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Adalimumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Golimumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Ustekinumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Certolizumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Adalimumab Golimumab Ustekinumab Certolizumab Tofacitinib Missing | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

<sup>&</sup>lt;sup>1</sup>Patients with intensification.

<sup>&</sup>lt;sup>2</sup>Patients with treatment discontinuation.

Patients with new biologic treatment.




Date: 17FEB2022

# Table 3.1.3 Follow-up

| Time of follow-up (months) n xx Mean (SD) Median (Q1, Q3) Min, Max Xx, xx Missing xx Xx.x (xx.x, xx.x) Xx.x (xx.x, xx | Median (O1 O3) | | | | |
|---|---|---|---|---|---|
| Median (Q1 Q3) | Median (Q1 Q3) | | | VDZ | Other Biologic |
| Median (Q1 Q3) | Median (Q1 Q3) | | | (n=xx) | (n=xx) |
| Median (Q1 Q3) | Median (Q1 Q3) | Time of follow-up (months) | n | xx | xx |
| Median (Q1, Q3) | Median (Q1, Q3) | | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Min, Max xx, xx Missing xx M | Missing xx Applies xx Missing by the Applies on Wand Subject to the Applies of Wand Subject to the Applies of Wand Subject | | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Missing xx ARP xx | Missing xx Appli xx Amarcial Use Only and Subject to the Appli xx | | Min, Max | xx, xx | xx xx |
| I JSE ONLY and Subject to the | omercial Use Only and Subject to the Principal | | Missing | xx | robj. xx |
| Jse Only and Subject to the | omercial Use Only and Subject to the | | Missing | XX | XX XX |
| | amercial | | 1126 OUTA | | |
| Colli | | ,40, | | | |
| * Hour Cour, | * 40. | .40, | | | |
| · For Hour Cour. | · kot Ho. | 1699. | | | |
| Leda: For Non-Con. | rega. For Ho. | · Kake | | | |
| E Lakeda: For Mon. Com. | ELakeda: For Ho. | 70, | | | |
| Jof Takedai. For Non. Com. | John Stephen S | | | | |
| Stor Takedai. For Non. Com. | of Takeda. For No. | | | | |
| of Takeda. For Won. Com. | ed of Takeda. For No. | | | | |
| of Takeda. For Non-Con. | of Takeda. For No. | | | | |
| y of Takeda. For Non-Con. | y of Takeda. For No. | | | | |



Study : EVOLVE

Date: 17FEB2022


**Table 3.1.4 Concomitant treatment** 

| | | VDZ | Other Biologic |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Any concomitant medication | during | | |
| induction | | | |
| Total no-missing | n | xx | xx © |
| No | n (%) | xx ( xx.x%) | xx (_xx.x%) |
| Yes* | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Corticosteroids | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Immunomodulators | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Antibiotics | n (%) | xx ( xx-x%) | xx ( xx.x%) |
| 5 – ASA | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Others | n (%) n (%) n during | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | A, xx | xx |
| | C | | |
| Any concomitant medication | during | | |
| maintenance | | | |
| Total no-missing | RIC. | xx | xx |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes* | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Corticosteroids | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Immunomoduators | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Antibiotics | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 5-ASA | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Others | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

<sup>\*</sup> More than an answer possible.



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

# 9.3.2 By treatment (CD patients)

# Table 3.2.1 Biologic index treatment I (CD patients)

| | • | · · · / | |
|---------------------------------------|-------|-------------|----------------|
| | | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) |
| Steroid status at index date | | | 1 Oly |
| Total no-missing | n | xx | xx Ø |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | iect | |
| · | · | . ( ) ) | · |

Table 3.3.1 Biologic index treatment I (CD-VDZ patients)

| | ie | | |
|---|---|---|---|
| | (OD VDZ | and Subject | |
| 9.3.3 By treatment line | (CD-VDZ patients) | | |
| | 50 | | |
| Table 3.3 | .1 Biologic index treatm | nent I (CD-VDZ patient | ts) |
| | Clo | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
| | we. | (n=xx) | (n=xx) |
| Steroid status at index date | 2111 | | |
| Total no-missing | n | xx | xx |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| O. | | | |



| Study : EVOLVE |
|----------------|

Date: 17FEB2022

# 9.3.4 By treatment line (CD-Other Biologic Patients)

Table 3.4.1 Biologic index treatment I (CD-Other Biologic patients)

| | | 1 <sup>st</sup> line | 2 <sup>nd</sup> line<br>(n=xx) |
|---|---|---|---|
| | | (n=xx) | |
| Steroid status at index date | | | \Q <sub>1</sub> |
| Total no-missing | n | xx | ··· C& Ole |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | CIJO | |
| | | 6, | |
| | | Agua | |
| | | 3 | |

# 9.3.5 By treatment (UC patients)

Table 3.5.1 Biologic index treatment I (UC patients)

| | ocicio. | VDZ | Other Biologic |
|------------------------------|---------|-------------|----------------|
| | Me. | (n=xx) | (n=xx) |
| Steroid status at index date | | | |
| Total no-missing | n | xx | xx |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| <br>O. | | | |


## 9.3.6 By treatment line (UC-VDZ patients)

Table 3.6.1 Biologic index treatment I (UC-VDZ patients)

| | | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Steroid status at index date | | | 10 |
| Total no-missing | n | xx | · C&O |
| Intolerant | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Dependent | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Refractory | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| None of the above | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | CILOI | |

# 9.3.7 By treatment line (UC-Other Biologic Patients)

Table 3.7.1 Biologic index treatment I (UC-Other Biologic patients)

| ame. | 1 <sup>st</sup> line | 2 <sup>nd</sup> line |
|---|---|---|
| | (n=xx) | (n=xx) |
| n | xx | xx |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%)<br>n (%)<br>n (%) | n xx n (%) xx (xx.x%) n (%) xx (xx.x%) n (%) xx (xx.x%) |

. . .



# 9.4 Primary objective (Endpoint analysis)

## 9.4.1 PS-IPTW

Table 4.1.1 Descriptive analysis pre and post PS-IPTW (CD patients)

| | | ٠. ٥ | Pre PS-IPTW | | Post PS-IPTW | |
|---|---|---|---|---|---|---|
| | | Subje | VDZ | Other Biologic | VDZ | Other Biologic |
| | | 79 | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | Ä | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Male<br>Female | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever CD diagnosis and index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | Never smoked | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| HBI overall score | 70 | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Perianal disease at diagnosis | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| HBI overall score Perianal disease at diagnosis Previous abdominal surgeries | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




Study : EVOLVE


Date: 17FEB2022

| | | _ | Pre PS-IPTW | | Post | PS-IPTW |
|---|---|---|---|---|---|---|
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous perianal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis | lleal | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Colonic/Ileocolonic | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Stricturing/Penetrating | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Treatment line | First biologic (bionaive) | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Second biologic | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Corticosteroids treatment administered within the 6 | Yes office | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| months prior the index date | .00 | | | | | |
| | L. College | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the 6 | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| months prior the index date | | | | | | |
| months prior the index date PCR (mg/L)[LOG] | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |



| | | Pro | Pre PS-IPTW | | PS-IPTW |
|---|---|---|---|---|---|
| | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Fecal calprotectin (mg/Kg)[LOG] | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within the Yes 6 months prior the index date? | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

Figure 4.1.1 Density Plot - pre PS-IPTW (CD)

Figure 4.1.2 Density Plot - Post-IPTW (CD)

Figure 4.1.3 Love Plot (CD)

Figure 4.1.4 Box Plots (CD)



| | | | | | | Date : 17FEB2022 |
|---|---|---|---|---|---|---|
| Table | 4.1.2 Descriptive analysis pre and | post PS-IPT | ·W (UC patie | ents)-2010 | | |
| | · · · | | | PS-IPTW | Post | t PS-IPTW |
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Female | h (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever UC diagnosis and index date (years) | Never smoked | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | Never smoked | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Partial Mayo score | alue. | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis | Proctitis/proctosigmoiditis / Left-sided | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| ×9. | Extensive colitis | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis Treatment line | First biologic (bionaive) | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| × 7.0 | Second biologic | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |



Study : EVOLVE


Date: 17FEB2022

| | | | Pre F | Pre PS-IPTW | | PS-IPTW |
|---|---|---|---|---|---|---|
| | | | VDZ | VDZ Other Biologic | | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Any Corticosteroids treatment administered within the 6 months prior the index date | Yes | n (%) | xxx (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the 6 months prior the index date | Yes | | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | | n (%) Mean (SE) Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Fecal calprotectin (mg/Kg)[LOG] | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within the 6 months prior the index date? | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

Figure 4.1.5 Density Plot – pre PS-IPTW (UC)

Figure 4.1.6 Density Plot - Post-IPTW (UC)

Figure 4.1.7 Love Plot (UC) hir Figure 4.1.8 Box Plots (UC) hir for water and some and the figure 4.1.8 box Plots (UC) hir for water and the figur All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II


| | | Study: EVOLVE |
|----------|---------------------------|------------------|
| | STATISTICAL ANALYSIS PLAN | Version : 6.0 |
| BIWLEVER | | Date : 17FEB2022 |

| | | | | 2.0 | 03 | Date : 17FEB2022 |
|---|---|---|---|---|---|---|
| Table 4 | 4.1.3 Descriptive analysis pre a | nd post PS-IPTW( | CD patients - | - First (Ine) | • | |
| | | | Pre I | Pre RS-IPTW Pos | | |
| | | | VDZ Ø | Other Biologic | VDZ | Other Biologic |
| | | | (n∋xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Female | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever CD diagnosis and index date ( | years) | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | Never smoked Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| HBI overall score | alhe | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Perianal disease at diagnosis | Yes CO | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Yes Correction Yes No Yes No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| × | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous perianal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| £ 7.0 | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |




Study : EVOLVE


Date: 17FEB2022

| | | | Pre PS-IPTW | | Post | PS-IPTW |
|---|---|---|---|---|---|---|
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Location of intestinal involvement at diagnosis | lleal | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Colonic/Ileocolonic | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Stricturing/Penetrating | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Corticosteroids treatment administered within the 6 months prior the index date | Yes No Yes No | 0(%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the 6 months prior the index date | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No OFFE | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | COM | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Fecal calprotectin (mg/Kg)[LOG] | Onto | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within the | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 6 months prior the index date? | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |



Figure 4.1.9 Density Plot - pre PS-IPTW (CD - First line)

Figure 4.1.10 Density Plot - Post-IPTW (CD - First line)

Jure 4.1.11 Love Plot (CD – First II).

Figure 4.1.12 Box Plots (CD – First line) All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



Table 4.1.4 Descriptive analysis pre and post PS-IPTW (UC patients – First line)

| | | | Pre PS-IPTW | | Post PS-IPTW | |
|---|---|---|---|---|---|---|
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Female | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever UC diagnosis and index date (years) | Never smoked | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | Never smoked | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Partial Mayo score | Current smoker Yes | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis | Proctitis/proctosigmoiditis / Left-sided | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 169'a. | Extensive colitis | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

SOPs ST 1008-06-II - CONFIDENTIAL- 



Study : EVOLVE


Date: 17FEB2022

| | | | | Pre Ps | S-IPTW | Post PS-IPTW | |
|---|---|---|---|---|---|---|---|
| | | | | VDZ Other Biologic | | VDZ | Other Biologic |
| | | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Any Corticosteroids treatment administered within the 6 | Yes | | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| months prior the index date | | | 3 | ,40 | | | |
| | No | | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the | Yes | | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 6 months prior the index date | | | n (%) | | | | |
| | No | 440 | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | | 0/, | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Fecal calprotectin (mg/Kg)[LOG] | | amercial Use Only? | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within | Yes | icial . | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| the 6 months prior the index date? | | dela | | | | | |
| | No | Oldi. | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |



Figure 4.1.13 Density Plot – pre PS-IPTW (UC – First line)

Figure 4.1.14 Density Plot – Post-IPTW (UC – First line)

Jensity Plot - Postigure 4.1.15 Love Plot (UC - First line)

Figure 4.1.16 Box Plots (UC - First line)

Figure 4.1.16 Box Plots (UC - First line) All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II

| | Study : EVOLVE |
|---------|------------------|
| BIWLEVE | Date : 17FEB2022 |

| | | | | | 703 | Date : 17FEB2022 |
|---|---|---|---|---|---|---|
| Table 4 | .1.5 Descriptive analysis pre an | d post PS-IPTW (C | D patients – | Second line) | • | |
| | . , , | · | Pre PS-IPTW Post PS-IPTW | | | |
| | | | VDZ Ø | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Female | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever CD diagnosis and index date | (years) | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | (years) Never smoked Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| HBI overall score | anne | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Perianal disease at diagnosis | Yes CO | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries Previous perianal surgeries | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous perianal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| X 10 | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |




Study : EVOLVE


Date: 17FEB2022

| | | _ | Pre PS-IPTW | | Post | PS-IPTW |
|---|---|---|---|---|---|---|
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Location of intestinal involvement at diagnosis | lleal | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Colonic/Ileocolonic | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Stricturing/Penetrating | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Corticosteroids treatment administered within the 6 | Yes No Yes No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| months prior the index date | Oly | ) | | | | |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the 6 | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| months prior the index date | *C,O | | | | | |
| | No No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | COLL | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Fecal calprotectin (mg/Kg)[LOG] | 10Pr | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within the | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 6 months prior the index date? | | | | | | |
| 6 months prior the index date? | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Reason for discontinuation (First line) | Primary failure | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

| | | <i>O</i> <sub>1</sub> |
|-------------|---------------------------|-----------------------|
| | | Study: EVOLVE |
| 71001011015 | STATISTICAL ANALYSIS PLAN | Version : 6.0 |
| Bl@Lever | | Date : 17FEB2022 |

| | | Pre F | Pre PS-IPTW | | PS-IPTW |
|---|---|---|---|---|---|
| | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Secondary failure | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Safety | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Other | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |

Figure 4.1.17 Density Plot – pre PS-IPTW (CD – Second line)

Jure 4.1.19 Love Plot (CD – Second I.

Figure 4.1.20 Box Plots (CD – Second line) Figure 4.1.18 Density Plot - Post-IPTW (CD - Second line)



| Table 4.1.6 Descriptive analysis pre and post PS-IPTW (UC patients – Second line) | | | | | | |
|---|---|---|---|---|---|---|
| | | | Pre | PS-IPTW | Post | PS-IPTW |
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Age at index date (years) | | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Sex | Male | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Female | h(%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Time between first ever UC diagnosis and index (years) | date Never smoked | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Smoking status at index treatment initiation | Never smoked | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Former smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Partial Mayo score | CORNI | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Previous abdominal surgeries | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | Current smoker Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis | Dura ditti da manda alima alilitis di la finalida di | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Location of intestinal involvement at diagnosis | Extensive colitis | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |




Study : EVOLVE


Date: 17FEB2022

| | | | Pre PS-IPTW | | Post PS-IPTW | |
|---|---|---|---|---|---|---|
| | | | VDZ | Other Biologic | VDZ | Other Biologic |
| | | | (n=xx) | (n=xx) | (n=xx) | (n=xx) |
| Any Corticosteroids treatment administered within the 6 months prior the index date | Yes | n (%) | xxix (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Any Immunomodulators treatment administered within the 6 months prior the index date | Yes | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| PCR (mg/L)[LOG] | OKK | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Fecal calprotectin (mg/Kg)[LOG] | USE | Mean (SE) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| The patient has had extra intestinal manifestation within the 6 months prior the index date? | Yes MRErcial Use Only | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| | No OFFIFT | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| Reason for discontinuation (First line) | Primary failure | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| d. | Secondary failure | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 80. | Safety | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |
| 80. | Other | n (%) | xx.x (xx.x) | xx.xx (xx.x) | xx.x (xx.x) | xx.xx (xx.x) |



Figure 4.1.21 Density Plot – pre PS-IPTW (UC – Second line)

Figure 4.1.22 Density Plot – Post-IPTW (UC – Second line)

Figure 4.1.23 Love Plot (UC - Second line)

Figure 4.1.24 Box Plots (UC - Second line)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



## 9.4.2 Discontinuation

**Table 4.2.1 Discontinuation** 

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with discontinuation | Total no-missing | Patients with | | |
| | n | n(%) | n n | n(%) | OR (IC95%)* | p-value* |
| CD | | 1 3170 | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Ileal Vs. VDZ – Colonic/Ileocolonic¹ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | Sex isla | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – Intensification Vs. VDZ – Colonic/Ileocolonic – ntesification¹ | MILLEXX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| /DZ – Ileal – No Intensification Vs. VDZ – Colonic/Ileocolonic – No ntesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ - 2 years or more diagnosis Vs. VDZ - less than 2 years liagnosis <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – 2 years or more diagnosis – 1 <sup>st</sup> line Vs. VDZ – less than 2 years liagnosis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II




Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gı | oup | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with discontinuation | Total no-missing | Patients with discontinuation | | |
| | n | n(%) | n ve | n(%) | OR (IC95%)* | p-value* |
| $DZ-2$ years or more diagnosis $-2^{nd}$ line Vs. $VDZ-$ less than 2 ears diagnosis $-2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | × × O | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx | xx ( xx.x%) | JOJ XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| DZ – Inflamatory – 1 <sup>st</sup> line Vs. VDZ – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – Inflamatory – 2 <sup>nd</sup> line Vs. VDZ – Stricturing/Penetrating – 2 <sup>nd</sup> | xx | xx.(-xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx c | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx S | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | AULT, XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Ileal – Intensification Vs. O.B. – Colonic/Ileocolonic – tesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| B. – Ileal – No Intensification Vs. O.B. – Colonic/Ileocolonic – No tesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B 2 years or more diagnosis Vs. O.B less than 2 years | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

diagnosis1



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gr | oup O | | |
|---|---|---|---|---|---|---|
| | | Patients with | | Patients with | | |
| | Total no-missing | discontinuation | Total no-missing | discontinuation | | |
| | n | n(%) | n 🗸 | n(%) | OR (IC95%)* | p-value* |
| O.B. $-2$ years or more diagnosis $-1^{st}$ line Vs. O.B. $-$ less than 2 years diagnosis $1^{st}$ line <sup>1</sup> | xx | xx ( xx.x%) | xx.O | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-2^{nd}$ line Vs. O.B. $-$ less than 2 years diagnosis $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | Propries | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx \sqrt{9} | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>2</sup> | ne <sup>xi</sup> ial | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> | MILL XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic <sup>2</sup> | XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic 1 <sup>st</sup> ine <sup>3</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> ( | group | | |
|---|---|---|---|---|---|---|
| | | Patients with | | Patients with | | |
| | Total no-missing | discontinuation | Total no-missing | discontinuation | | |
| | n | n(%) | n Ne | n(%) | OR (IC95%)* | p-value* |
| VDZ – Ileal Vs. O.B. – Ileal² | xx | xx ( xx.x%) | XXO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | S xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | ) xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years | XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis <sup>2</sup> | | ouly. | | | | |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| years diagnosis – 1 <sup>st</sup> line <sup>3</sup> | 1)9 | | | | | |
| $VDZ$ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| years diagnosis – 2 <sup>nd</sup> line <sup>4</sup> | Willek Cigil | | | | | |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis <sup>2</sup> | Oll | | | | | |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis – 1 <sup>st</sup> line <sup>3</sup> | | | | | | |
| VDZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis – 2 <sup>nd</sup> line⁴ | | | | | | |
| /DZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

| | <i>Q</i> <sub>1</sub> |
|---------|-----------------------|
| | Study : EVOLVE |
| BIWLEVE | Date : 17FEB2022 |

| | 1 <sup>st</sup> gı | roup | 2 <sup>nd</sup> gro | oup Jole | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with discontinuation | Total no-missing | Patients with discontinuation | | |
| | n | n(%) | n Ne | n(%) | OR (IC95%)* | p-value* |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Inflamatory – 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-Inflamatory-2^{nd}\ line\ Vs.\ O.BInflamatory-2^{nd}\ line\ ^4$ | XX | xx ( xx.x%) | XX XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating <sup>2</sup> | xx | xx ( xx.x%) | ) xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating $-1^{st}$ line Vs. O.B. $-$ Stricturing/Penetrating $-1^{st}$ line $^3$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating – $2^{\rm nd}$ line Vs. O.B. – Stricturing/Penetrating – $2^{\rm nd}$ line $^4$ | xx xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| uc | ial | | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | Sxx . | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis¹ | Mill xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ$ – Extensive colitis – $2^{nd}$ line $Vs.$ $VDZ$ – $Proctitis/Left$ colitis – $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – Intensification Vs. VDZ – Proctitis/Left colitis – Intesification¹ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with discontinuation | Total no-missing | Patients with discontinuation | | |
| | n | n(%) | n ve | n(%) | OR (IC95%)* | p-value* |
| /DZ – Extensive colitis – No Intensification Vs. VDZ – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xxO xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ - 2 years or more diagnosis Vs. $VDZ - less$ than 2 years agnosis <sup>1</sup> | xx | xx ( xx.x%) | Original xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| DZ - 2 years or more diagnosis $-1$ <sup>st</sup> line Vs. VDZ $-$ less than 2 years agnosis $-1$ <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| $DZ-2$ years or more diagnosis $-2^{nd}$ line Vs. $VDZ-$ less than 2 ears diagnosis $-2^{nd}$ line <sup>1</sup> | xx \S | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| .B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xxi (2) | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | Wexx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis – 1 <sup>st</sup> | offi, xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis = 2 <sup>nd</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| .B. – Extensive colitis – Intensification Vs. O.B. – Proctitis/Left colitis | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

Intesification<sup>1</sup>



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gro | oup Jole | | |
|---|---|---|---|---|---|---|
| | Total no missing | Patients with | Total na missina | Patients with | | |
| | Total no-missing | discontinuation n(%) | Total no-missing n | discontinuation n(%) | OR (IC95%)* | p-value* |
| D.B. – Extensive colitis – No Intensification Vs. O.B. – Proctitis/Left olitis – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| D.B 2 years or more diagnosis Vs. O.B less than 2 years liagnosis <sup>1</sup> | xx | xx ( xx.x%) | Ollo xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| D.B. – 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years iagnosis 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $0.B2$ years or more diagnosis $-2^{nd}$ line Vs. $0.B$ less than 2 ears diagnosis $2^{nd}$ line <sup>1</sup> | xx \sqrt{9} | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ Vs. O.B. <sup>5</sup> | Julius xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> | Wexx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis⁵ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> ne <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> ine <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gı | roup | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with discontinuation | Total no-missing | Patients with discontinuation | | |
| | n | n(%) | n we | n(%) | OR (IC95%)* | p-value* |
| VDZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | XX XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ$ – Extensive colitis – $2^{nd}$ line Vs. O.B. – Extensive colitis – $2^{nd}$ line <sup>7</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ$ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>7</sup> | ALIMERCIAL XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis <sup>5</sup> | OMMEXX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more diagnosis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more diagnosis – 2 <sup>nd</sup> line <sup>7</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

<sup>\*</sup>Estimated with a logistic regression

<sup>&</sup>lt;sup>1</sup>Data without PS-IPTW.



<sup>2</sup>Data with PS-IPTW (CD).

<sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).

<sup>5</sup>Data with PS-IPTW (UC).

<sup>6</sup>Data with PS-IPTW (UC-1<sup>st</sup> line).

<sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II

| | , 150 | Study : EVOLVE |
|----------|-------|------------------|
| BIWLEVER | MS. | Date : 17FEB2022 |

Table 4.2.2 CD patients with VDZ – Discontinuation Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| flodel | xx | xx xx | |
| ine treatment | × ×0 | | x.xxxx |
| /pe of diagnosis | 79/8CL | | x.xxxx |
| isease duration | , SUIV. | | x.xxxx |
| ype of disease behaviour at diagnosis | allo | | x.xxxx |
| nteraction Line treatment and Type of diagnosis | 4 | | x.xxxx |
| teraction Line treatment and Disease duration teraction Line treatment and Type of disease behaviour at diagnosis teraction Type of diagnosis and Disease duration | | | x.xxxx |
| teraction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Type of diagnosis and Disease duration | | | x.xxxx |
| teraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Disease duration | | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |


| | Study : EVOLVE |
|----------|------------------|
| Bl@Lever | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | dico | X.XXXX |

Table 4.2.3 CD patients with VDZ - Discontinuation Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | 15 <sup>©</sup> | |
| 2 <sup>nd</sup> line | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line<br> | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |

Note: Only significant variables and/or interactions (Table 4.1.3) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | <i>Q</i> <sub>1</sub> |
|---------|-----------------------|
| | Study: EVOLVE |
| Blocker | Date : 17FEB2022 |

Table 4.2.4 UC patients with VDZ – Discontinuation Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | xx xx | |
| Line treatment | , | ,00 | x.xxxx |
| Type of diagnosis | iec | | x.xxxx |
| Disease duration | Subjec | | x.xxxx |
| Interaction Line treatment and Type of diagnosis | and | | x.xxxx |
| Interaction Line treatment and Disease duration | KING | | x.xxxx |
| Interaction Type of diagnosis and Disease duration | °⊗<br>O, | | x.xxxx |
| Interaction Line treatment, Type of diagnosis and Disease duration | 1/2 | | x.xxxx |


| | | | Study : EVOLVE |
|----------|---------------------------|----|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | MS | Date : 17FEB2022 |

Table 4.2.5 UC patients with VDZ – Discontinuation Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Subjection | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| | O' | |

Note: Only significant variables and/or interactions (Table 4.1.3) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | | | Study : EVOLVE |
|----------|---------------------------|---|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | K | Date : 17FEB2022 |

| | | Me Lo. | |
|---|---|---|---|
| Table 4.2.6 CD patients with Other Biologic – Discontin | nuation Logistic | regression model (p-values | ) |
| | n | Missing | p-value |
| del | xx | **/© xx | |
| e treatment | . * | 0 | x.xxxx |
| pe of diagnosis | 196Cr | | x.xxxx |
| sease duration | enly, | | x.xxxx |
| pe of disease behaviour at diagnosis | and | | x.xxxx |
| del e treatment pe of diagnosis ease duration pe of disease behaviour at diagnosis eraction Line treatment and Type of diagnosis eraction Line treatment and Disease duration eraction Line treatment and Type of disease behaviour at diagnosis eraction Type of diagnosis and Disease duration eraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Line treatment and Disease duration | | | x.xxxx |
| eraction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Line treatment, Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| raction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |


| | Study: EVOLVE |
|----------|------------------|
| Bl@Lever | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | dico | X.XXXX |

Table 4.2.7 CD patients with Other Biologic – Discontinuation Logistic regression model (estimated OR)

| | *** | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | 2nd line Vs. 1st line Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Se | |
| 2 <sup>nd</sup> line | lleal Vs. Colonic/lleocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | lleal Vs. Colonic/lleocolonic | xx.x (xx.x, xx.x) |
| | alle | |

Note: Only significant variables and/or interactions (Table 4.1.3) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | | | Study : EVOLVE |
|----------|---------------------------|---|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | K | Date : 17FEB2022 |

Table 4.2.8 UC patients with Other Biologic - Discontinuation Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | xx xx | |
| ine treatment | | **0 | x.xxxx |
| ype of diagnosis | Sil | e <sub>Cr</sub> | x.xxxx |
| Disease duration | Sul | ) > | x.xxxx |
| nteraction Line treatment and Type of diagnosis | and | | x.xxxx |
| nteraction Line treatment and Disease duration | ally | | x.xxxx |
| nteraction Type of diagnosis and Disease duration | ۯ, | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Disease duration | 173 | | x.xxxx |

| | <i>Q</i> <sub>1</sub> |
|---------|-----------------------|
| | Study : EVOLVE |
| Blocker | Date : 17FEB2022 |

Table 4.2.9 UC patients with Other Biologic - Discontinuation Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Subjection | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |

Note: Only significant variables and/or interactions (Table 4.1.3) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.



# 9.4.3 Time to treatment discontinuation

Table 4.3.1 Time to treatment discontinuation (Months)

| | 1 <sup>st</sup> group 2 <sup>nd</sup> group | | | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment discontinuation** Median(Q1,Q3) | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | p-value*** |
| CD | | CUDIO | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. VDZ – Colonic/Ileocolonic¹ | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx O <sub>L</sub> | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | New Contraction of the Contracti | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – Intensification Vs. VDZ – Colonic/Ileocolonic – Intesification <sup>1</sup> | xx x | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – No Intensification Vs. VDZ – Colonic/Ileocolonic – No Intesification <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-2$ years or more diagnosis – $1^{st}$ line $Vs.\ VDZ-$ less than 2 years diagnosis – $1^{st}$ line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $ 2^{\text{nd}}$ line Vs, VDZ $-$ less than 2 years diagnosis $ 2^{\text{nd}}$ line $^{\text{1}}$ | xx | xx.x (xx.x, xx.x) | хх | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | <b>2</b> <sup>rrd</sup> 9 | )<br> roup | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment discontinuation** Median(Q1,Q3) | p-value*** |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. VDZ – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | *Ke xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. VDZ – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | xx Oul | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – Intensification Vs. O.B. – Colonic/Ileocolonic – Intesification <sup>1</sup> | SX. | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – No Intensification Vs. O.B. – Colonic/Ileocolonic – No Intesification <sup>1</sup> | icial xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 1 <sup>st</sup> line Vs. O.B. $-$ less than 2 years diagnosis 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-2^{\rm nd}$ line Vs. O.B. $-$ less than 2 years diagnosis $2^{\rm nd}$ line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> ç | group | 2 <sup>nd</sup> ç | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | p-value*** |
| O.B. – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | */\omega_ xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Vs. O.B. <sup>2</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic 1 <sup>st</sup> line <sup>3</sup> | xx Orli | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic 2 <sup>nd</sup> line <sup>4</sup> | SX. | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. O.B. – Ileal² | | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | xx xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis² | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis – 1 <sup>st</sup> line <sup>3</sup> | | | | | |
| VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ - 2 years or more diagnosis Vs. O.B 2 years or more diagnosis <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> group | | 2 <sup>nd</sup> c | 2 <sup>nd</sup> group | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | p-value*** |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more diagnosis – 1 <sup>st</sup> line <sup>3</sup> | хх | xx.x (xx.x, xx.x) | Silvo xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $2^{\text{nd}}$ line Vs. O.B. – 2 years or more diagnosis – $2^{\text{nd}}$ line $^4$ | xx | xx.x (xx.x, xx,x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Inflamatory – 1 <sup>st</sup> line <sup>3</sup> | xx 🔏 | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Inflamatory – 2 <sup>nd</sup> line <sup>4</sup> | xx Olym | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating <sup>2</sup> | XX C | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Stricturing/Penetrating $-1^{st}$ line Vs. O.B. $-$ Stricturing/Penetrating $-1^{st}$ line $^3$ | Ki XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating – 2 <sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>4</sup> | хх | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| UC VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> ( | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | p-value*** |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | the xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis – Intensification Vs. VDZ – Proctitis/Left colitis – Intesification <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – No Intensification Vs. VDZ – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx 🚜 | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $-$ 1st line Vs. VDZ $-$ less than 2 years diagnosis $-$ 1st line 1 | xx Offi | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 2 <sup>nd</sup> line <sup>1</sup> | id xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – Intensification Vs. O.B. – Proctitis/Left colitis – Intesification <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> 9 | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | p-value*** |
| O.B. – Extensive colitis – No Intensification Vs. O.B. – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx | xx.x (xx.x, xx.x) | THE XX | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B 2 years or more diagnosis - 1 <sup>st</sup> line Vs. O.B less than 2 years diagnosis 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. O.B. $-$ less than 2 years diagnosis 2 <sup>nd</sup> line <sup>1</sup> | xx orly | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>5</sup> | w <sup>©</sup> | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> | xx xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> line <sup>6</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Extensive colitis – 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> group | | <b>2</b> <sup>rrd</sup> g | 2 <sup>rd</sup> group | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n | Time to treatment<br>discontinuation**<br>Median(Q1,Q3) | Total no-missing* | Time to treatment discontinuation** Median(Q1,Q3) | p-value*** |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | XX | xx.x (xx.x, xx.x) | *// <sub>©</sub> xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis – $1^{st}$ line $^6$ VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line $^7$ | xx | xx.x(xx-x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. − 2 years or more diagnosis <sup>5</sup> | xx 🕠 | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more diagnosis | xx Olum | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| - 1 <sup>st</sup> line <sup>6</sup> | 150 | | | | |
| VDZ - 2 years or more diagnosis – $2^{\text{nd}}$ line Vs. O.B. – 2 years or more diagnosis – $2^{\text{nd}}$ line $^7$ | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |

<sup>\*</sup> Patients with correct data to calculate "time to treatment discontinuation".

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II


<sup>\*\*</sup> Estimated with Kaplan-Meier method.

<sup>\*\*\*</sup> Estimated with LogRank test.

<sup>&</sup>lt;sup>1</sup>Data without PS-IPTW.

<sup>&</sup>lt;sup>2</sup>Data with PS-IPTW (CD).

<sup>&</sup>lt;sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>&</sup>lt;sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).

<sup>&</sup>lt;sup>5</sup>Data with PS-IPTW (UC).



<sup>6</sup>Data with PS-IPTW (UC-1st line).

<sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



# 9.4.4 Duration of treatment

**Table 4.4.1 Duration of treatment (Months)** 

| | 1 <sup>st</sup> group 2 <sup>nd</sup> group | | | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| CD | | Culoje | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. VDZ – Colonic/Ileocolonic¹ | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx - xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – Intensification Vs. VDZ – Colonic/Ileocolonic – Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – No Intensification Vs. VDZ – Colonic/Ileocolonic – No Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $-$ 1 <sup>st</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis - 2 <sup>nd</sup> line Vs. VDZ - less than 2 years diagnosis - 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2nd gi | roup | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. VDZ – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | *Ko xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. VDZ – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | ×× | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – Intensification Vs. O.B. – Colonic/Ileocolonic – Intesification <sup>1</sup> | xx (xx - xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – No Intensification Vs. O.B. – Colonic/Ileocolonic – No Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 1 <sup>st</sup> line Vs. O.B. $-$ less than 2 years diagnosis 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-2^{\rm nd}$ line Vs. O.B. $-1$ less than 2 years diagnosis $2^{\rm nd}$ line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | roup | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing* | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| O.B. – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | *Ko xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>2</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic² | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic 1 <sup>st</sup> line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-Colonic/Ileocolonic-2^{nd}\ line\ Vs.\ O.BColonic/Ileocolonic\ 2^{nd}\ line^4$ | xx (xx-xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal Vs. O.B. – Ileal² | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis² | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – less than 2 years diagnosis – $1^{st}$ line Vs. O.B. – less than 2 years diagnosis – $1^{st}$ line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 2 <sup>nd</sup> line Vs. O.B. – less than 2 years diagnosis – 2 <sup>nd</sup> line <sup>4</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B2 years or more diagnosis <sup>2</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gı | oup | 2nd gi | oup | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing*<br>n (n₁ - n₂) | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| VDZ - 2 years or more diagnosis – $1^{st}$ line Vs. O.B. – 2 years or more diagnosis – $1^{st}$ line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | SHO XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $$ - 2 years or more diagnosis – $2^{nd}$ line Vs. O.B. – 2 years or more diagnosis – $2^{nd}$ line $^4$ | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Inflamatory – 1 <sup>st</sup> line <sup>3</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Inflamatory – 2 <sup>nd</sup> line <sup>4</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating <sup>2</sup> | xx (xx - xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating $-$ 1 <sup>st</sup> line Vs. O.B. $-$ Stricturing/Penetrating $-$ 1 <sup>st</sup> line $^3$ | (xx - xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating – $2^{\rm nd}$ line Vs. O.B. – Stricturing/Penetrating – $2^{\rm nd}$ line $^4$ | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| nc Toll, | | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis | xx(xx-xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | o<br>roup | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing* | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | *KLO XX | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – Extensive colitis – Intensification Vs. VDZ – Proctitis/Left colitis – Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – No Intensification Vs. VDZ – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ-2 years or more diagnosis – 1 <sup>st</sup> line Vs. $VDZ$ – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis—1 <sup>st</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – Intensification Vs. O.B. – Proctitis/Left colitis – Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing* | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| O.B. – Extensive colitis – No Intensification Vs. O.B. – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | illo, xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx(xx - xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 1st line Vs. O.B. $-$ less than 2 years diagnosis 1st line $^{1}$ | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. O.B. $-$ less than 2 years diagnosis $2^{nd}$ line <sup>1</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>5</sup> | xx (xx - xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis <sup>5</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> line <sup>6</sup> | xx(xx-xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> line <sup>7</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Extensive colitis – 2 <sup>nd</sup> line <sup>7</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



| Study : EVOLVE |
|----------------|

Date : 17FEB2022

| | 1 <sup>st</sup> gı | roup | 2 <sup>nd</sup> g | | |
|---|---|---|---|---|---|
| | Total no-missing*<br>n (n <sub>1</sub> - n <sub>2</sub> ) | Duration of<br>treatment**<br>Median(Q1,Q3) | Total no-missing* | Duration of<br>treatment**<br>Median(Q1,Q3) | p-value*** |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | the xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $1^{st}$ line Vs. O.B. – less than 2 years diagnosis – $1^{st}$ line $^6$ | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – less than 2 years diagnosis – $2^{\rm nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{\rm nd}$ line <sup>7</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis <sup>5</sup> | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more | xx (xx – xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis – $1^{st}$ line <sup>6</sup><br>VDZ - 2 years or more diagnosis – $2^{nd}$ line Vs. O.B. – 2 years or more diagnosis – $2^{nd}$ line <sup>7</sup> | (i xx (xx - xx) | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |

<sup>\*</sup>Patients with correct data to calculate "duration of treatment" n<sub>1</sub>: Patients treatment discontinued. n<sub>2</sub>: Patients treatment continue.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II


<sup>\*\*</sup>Estimated with Kaplan-Meier method.

<sup>\*\*\*</sup>LogRank test test.

<sup>&</sup>lt;sup>1</sup>Data without PS-IPTW.

<sup>&</sup>lt;sup>2</sup>Data with PS-IPTW (CD).

<sup>&</sup>lt;sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>&</sup>lt;sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line)

<sup>&</sup>lt;sup>5</sup>Data with PS-IPTW (UC).



<sup>6</sup>Data with PS-IPTW (UC-1<sup>st</sup> line).

Figure 4.4.1 Duration of treatment (months).

et's curves will presented.

Only and Subject to the control of t All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



# 9.4.5 Intensification

Table 4.5.1 Patients with one intensification or more (%)

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | group | | |
|---|---|---|---|---|---|---|
| | | Patients with one | *O | Patients with one | | |
| | | intensification or | cò. | intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) C | n | n(%) | OR (IC95%)* | p-value* |
| CD | | and | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx (xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. VDZ – Colonic/Ileocolonic <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | wildle xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – Intensification Vs. VDZ – Colonic/Ileocolonic – Intesification <sup>1</sup> | omittexx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – No Intensification Vs. VDZ – Colonic/Ileocolonic – No Intesification¹ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. VDZ - less than 2 years | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis <sup>1</sup> $VDZ - 2 \text{ years or more diagnosis} - 1^{\text{st}} \text{ line Vs. VDZ} - \text{less than 2 years}$ $\text{diagnosis} - 1^{\text{st}} \text{ line}^{1}$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | <i>O</i> 1 |
|----------|------------------|
| | Study : EVOLVE |
| BIOLEVER | Date : 17FEB2022 |

| | 1 <sup>st</sup> gr | oup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | | Patients with one | | Patients with one | | |
| | Total no-missing | intensification or more | Total no-missing | intensification or more | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| VDZ $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | , biecx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. VDZ – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. VDZ – Stricturing/Penetrating – 2 <sup>nd</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| line <sup>1</sup> | , 6 | 2 | | | | |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | MILL XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – Intensification Vs. O.B. – Colonic/Ileocolonic – | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| Intesification <sup>1</sup> O.B. – Ileal – No Intensification Vs. O.B. – Colonic/Ileocolonic – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II

| | <i>O</i> 1 |
|----------|------------------|
| | Study : EVOLVE |
| BIOLEVER | Date : 17FEB2022 |

| | 1 <sup>st</sup> gro | oup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | | Patients with one | | Patients with one | | |
| | Total no-missing | intensification or<br>more | Total no-missing | intensification or more | | |
| | _ | | ille | | OB (IC059/.)* | n vol* |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years | XX | xx ( xx.x%) | Cxx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis <sup>1</sup> | | | $\eta_0$ , | | | |
| O.B. $-2$ years or more diagnosis $-1$ <sup>st</sup> line Vs. O.B. $-$ less than 2 years diagnosis $1$ <sup>st</sup> line <sup>1</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis i line | | 31 | | | | |
| O.B. $-2$ years or more diagnosis $-2^{nd}$ line Vs. O.B. $-$ less than 2 years diagnosis $2^{nd}$ line <sup>1</sup> | XX | xx (xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| | 5 | <b>3</b> | | ( 0() | , | |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – $1^{st}$ line Vs. O.B. – Stricturing/Penetrating – $1^{st}$ line $1^{st}$ | weigh was | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| $O.BInflamatory-2^{nd}\ line\ Vs.\ O.BStricturing/Penetrating-2^{nd}$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| line <sup>1</sup> | | | | | | |
| VDZ Vs. O.B. <sup>2</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>2</sup> VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic <sup>2</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gro | oup | 2 <sup>nd</sup> g | group | | |
|---|---|---|---|---|---|---|
| | ı | Patients with one | | Patients with one | | |
| | i | intensification or | | intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| $\label{eq:VDZ-Colonic/Ileocolonic-1} VDZ-Colonic/Ileocolonic \ 1^{st} \ line^3$ $\ line^3$ | XX | xx ( xx.x%) | lojecx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $\label{eq:VDZ-Colonic/Ileocolonic-2nd} \mbox{VDZ-Colonic/Ileocolonic} \ 2^{\mbox{\scriptsize nd}} \ \mbox{line}^4$ $\mbox{line}^4$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. O.B. – Ileal² | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis² | Mexial | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>3</sup> | on xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis² | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gro | oup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | 1 | Patients with one | | Patients with one | | |
| | | intensification or | | intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| VDZ - 2 years or more diagnosis – $1^{st}$ line Vs. O.B. – 2 years or more diagnosis – $1^{st}$ line $^3$ | xx | xx ( xx.x%) | lipieci | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $2^{\text{nd}}$ line Vs. O.B. – 2 years or more diagnosis – $2^{\text{nd}}$ line $^4$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-Inflamatory-1^{st}\ line\ Vs.\ O.BInflamatory-1^{st}\ line\ ^3$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Inflamatory – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating $^2$ | xx in | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating $-$ 1 <sup>st</sup> line Vs. O.B. $-$ Stricturing/Penetrating $-$ 1 <sup>st</sup> line $^3$ | ORINAXX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Stricturing/Penetrating $-2^{\rm nd}$ line Vs. O.B. $-$ Stricturing/Penetrating $-2^{\rm nd}$ line $^4$ | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| UC VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | | | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gr | oup | 2 <sup>nd</sup> gr | roup | | |
|---|---|---|---|---|---|---|
| | | Patients with one | | Patients with one | | |
| | | intensification or | 4 | intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. $VDZ$ – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | Jojeck | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $\label{eq:VDZ-Extensive} VDZ-Extensive\ colitis-2^{nd}\ line\ Vs.\ VDZ-Proctitis/Left\ colitis-2^{nd}$ $line^1$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – Intensification Vs. VDZ – Proctitis/Left colitis – Intesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis – No Intensification Vs. VDZ – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx US | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ - 2 years or more diagnosis Vs. $VDZ$ - less than 2 years diagnosis <sup>1</sup> | MINEX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis – 1 <sup>st</sup> line Vs. VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis - $2^{nd}$ line Vs. VDZ - less than 2 years diagnosis - $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gro | oup | 2 <sup>nd</sup> g | proup 000 | | |
|---|---|---|---|---|---|---|
| | | Patients with one | | Patients with one | | |
| | | intensification or | Tatal na milaning | intensification or | | |
| | Total no-missing | more | Total no-missing | | OD (IO05%))* | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| $\label{eq:obs_equation} O.B Extensive \ colitis - 1^{st} \ line \ Vs. \ O.B Proctitis/Left \ colitis - 1^{st}$ | xx | xx ( xx.x%) | Cxx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| line <sup>1</sup> | | | 1101 | | | |
| O.B. – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis – 2 <sup>nd</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| line <sup>1</sup> | | Silve | | | | |
| O.B. – Extensive colitis – Intensification Vs. O.B. – Proctitis/Left colitis | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| - Intesification <sup>1</sup> | | O' | | | | |
| O.B. – Extensive colitis – No Intensification Vs. O.B. – Proctitis/Left | xx \S | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| colitis – No Intesification <sup>1</sup> | :0 | | | | | |
| O.B 2 years or more diagnosis Vs. O.B less than 2 years | xx J | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis <sup>1</sup> | allie | , | | , | , | |
| O.B. – 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| diagnosis 1 <sup>st</sup> line <sup>1</sup> | 70. | 701 (707.70) | ,,,, | 70t (70ti)/70 | your (round, round) | 7.000 |
| O.B. – 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – less than 2 | XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| years diagnosis 2 <sup>nd</sup> line <sup>1</sup> | ^^ | AA ( AA.A70) | ** | XX ( XX.X70) | ^^.^ (^^.^, ^^.^) | ۸.۸۸۸ |
| <i>☆</i> · | | ( 0( ) | | ()() | | |
| VDZ Vs. O.B. <sup>5</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gr | oup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | | Patients with one | | Patients with one | | |
| | | intensification or | | intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) | n n | n(%) | OR (IC95%)* | p-value* |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx | xx ( xx.x%) | Cxx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis <sup>5</sup> | XX | xx ( xx.x%) | ))) xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> line <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx 103 | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | XX XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Extensive colitis – 2 <sup>nd</sup> line <sup>7</sup> | MIN XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. 0.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> ( | proup proup | | |
|---|---|---|---|---|---|---|
| | | Patients with one intensification or | | Patients with one intensification or | | |
| | Total no-missing | more | Total no-missing | more | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis <sup>5</sup> | xx | xx ( xx.x%) | Jojeck | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $1^{\text{st}}$ line Vs. O.B. – 2 years or more diagnosis – $1^{\text{st}}$ line $^6$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $2^{nd}$ line Vs. O.B. – 2 years or more diagnosis – $2^{nd}$ line <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

<sup>\*</sup>Estimated with a logistic regression.

<sup>&</sup>lt;sup>1</sup>Data without PS-IPTW.

<sup>&</sup>lt;sup>2</sup>Data with PS-IPTW (CD).

<sup>&</sup>lt;sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>&</sup>lt;sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).

<sup>&</sup>lt;sup>5</sup>Data with PS-IPTW (UC).

<sup>&</sup>lt;sup>6</sup>Data with PS-IPTW (UC-1<sup>st</sup> line).

<sup>&</sup>lt;sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

| | | | Study : EVOLVE |
|----------|---------------------------|----|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | MS | Date : 17FEB2022 |

| | | | Date : 171 ED20 |
|---|---|---|---|
| | | 101 | |
| Table 4.5.2 CD patients with VDZ – One intensification | on or more Logistic | c regression model (p-value | s) |
| | n | Missing | p-value |
| pe of diagnosis sease duration pe of disease behaviour at diagnosis teraction Line treatment and Type of diagnosis teraction Line treatment and Disease duration teraction Line treatment and Type of disease behaviour at diagnosis teraction Type of diagnosis and Disease duration | xx | xx xx | |
| ne treatment | _ X | 0 | x.xxxx |
| pe of diagnosis | , iect | | x.xxxx |
| sease duration | SIID, | | x.xxxx |
| pe of disease behaviour at diagnosis | and | | x.xxxx |
| eraction Line treatment and Type of diagnosis | H | | x.xxxx |
| eraction Line treatment and Disease duration | | | x.xxxx |
| eraction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Line treatment, Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

| | Study: EVOLVE |
|----------|------------------|
| Blælever | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | dico | X.XXXX |

Table 4.5.3 CD patients with VDZ – One intensification or more Logistic regression model (estimated OR)

| | iect | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | | |
| 2 <sup>nd</sup> line | Ileal Vs. Colonic/lleocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| | Coz. | |

Note: Only significant variables and/or interactions (Table 4.4.2) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | <i>Q</i> <sub>1</sub> |
|---------|-----------------------|
| | Study: EVOLVE |
| Blocker | Date : 17FEB2022 |

Table 4.5.4 UC patients with VDZ - One intensification or more Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | **/© xx | |
| Line treatment | | ,00 | x.xxxx |
| Type of diagnosis | i,e <sup>C</sup> | | x.xxxx |
| Disease duration | Siloje | | x.xxxx |
| Interaction Line treatment and Type of diagnosis | and | | x.xxxx |
| Interaction Line treatment and Disease duration | KING | | x.xxxx |
| Interaction Type of diagnosis and Disease duration | °⊗<br>O, | | x.xxxx |
| Interaction Line treatment, Type of diagnosis and Disease duration | 1/2 | | x.xxxx |

| | | | Study : EVOLVE |
|----------|---------------------------|----|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | MS | Date : 17FEB2022 |

Table 4.5.5 UC patients with VDZ - One intensification or more Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Sul, | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |

Note: Only significant variables and/or interactions (Table 4.4.4) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | <i>Q</i> <sub>1</sub> |
|---------|-----------------------|
| | Study: EVOLVE |
| Blocker | Date : 17FEB2022 |

Table 4.5.6 CD patients with Other Biologic – One intensification or more Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | and Subject to W | & xx | |
| ine treatment | , 10 | * | x.xxxx |
| /pe of diagnosis | Niect. | | x.xxxx |
| isease duration | Sulvi | | x.xxxx |
| ype of disease behaviour at diagnosis | allo | | x.xxxx |
| nteraction Line treatment and Type of diagnosis | 3 | | x.xxxx |
| teraction Line treatment and Disease duration teraction Line treatment and Type of disease behaviour at diagnosis teraction Type of diagnosis and Disease duration | | | x.xxxx |
| steraction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Type of diagnosis and Disease duration | | | x.xxxx |
| iteraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Disease duration | | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| teraction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| steraction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | | Study: EVOLVE |
|-------------|---------------------------|------------------|
| DISOLON (OK | STATISTICAL ANALYSIS PLAN | Version : 6.0 |
| Bl@Lever | | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | Olico | X.XXXX |

Table 4.5.7 CD patients with Other Biologic – One intensification or more Logistic regression model (estimated OR)

| | iect | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | | |
| 2 <sup>nd</sup> line | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | lleal Vs. Colonic/lleocolonic | xx.x (xx.x, xx.x) |
| | Co | |

Note: Only significant variables and/or interactions (Table 4.4.2) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | <i>O</i> <sub>1</sub> |
|----------|-----------------------|
| | Study: EVOLVE |
| BIWLEVER | Date : 17FEB2022 |

Table 4.5.8 UC patients with Other Biologic – One intensification or more Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | xx xx | |
| Line treatment | | **0 | x.xxxx |
| Type of diagnosis | i e | | x.xxxx |
| Disease duration | Subje | | x.xxxx |
| Interaction Line treatment and Type of diagnosis | and | | x.xxxx |
| Interaction Line treatment and Disease duration | H | | x.xxxx |
| Interaction Type of diagnosis and Disease duration | Se Or | | x.xxxx |
| Interaction Line treatment, Type of diagnosis and Disease duration | 100 | | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | Study: EVOLVE |
|----------|------------------|
| Bl@Lever | Date : 17FEB2022 |

Table 4.5.9 UC patients with Other Biologic – One intensification or more Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Suble | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| | 81 | |

Note: Only significant variables and/or interactions (Table 4.4.4) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# 9.4.6 Time to first intensification

Table 4.6.1 Time to first intensification (Months)

| | 1 <sup>st</sup> group 2 <sup>nd</sup> gro | | | roup | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** | Total no-missing* | Time to first intensification** | |
| | n | Median(Q1,Q3) | n | Median(Q1,Q3) | p-value*** |
| CD | | Suble | | | |
| $VDZ - 1^{st}$ line $Vs. VDZ - 2^{nd}$ line <sup>1</sup> | xx | xx x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. VDZ – Colonic/Ileocolonic <sup>1</sup> | xx M | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx O | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | XX O | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx (S) | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis - 1 <sup>st</sup> line Vs. VDZ - less than 2 years diagnosis - 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. VDZ – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. VDZ – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | XX | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | roup | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** | Total no-missing* | Time to first intensification** | |
| | n | Median(Q1,Q3) | n | Median(Q1,Q3) | p-value*** |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | ille xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx | XX.X (XX.X, XX.X) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-$ 2 years or more diagnosis $-$ 1st line Vs. O.B. $-$ less than 2 years | xx OU | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis 1st line1 | 150 | | | | |
| O.B. $-$ 2 years or more diagnosis $-$ 2 <sup>nd</sup> line Vs. O.B. $-$ less than 2 years diagnosis $2^{\rm nd}$ line <sup>1</sup> | icial xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Stricturing/Penetrating – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic² | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>rd</sup> g | roup | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** Median(Q1,Q3) | Total no-missing* | Time to first intensification** Median(Q1,Q3) | p-value*** |
| VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic 1 <sup>st</sup> line <sup>3</sup> | xx | xx.x (xx.x, xx.x) | illo xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic 2 <sup>nd</sup> line <sup>4</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal Vs. O.B. – Ileal <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis² | xx Oly | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $1^{st}$ line Vs. O.B. – less than 2 years diagnosis – $1^{st}$ line <sup>3</sup> | Nasc . | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| $VDZ$ – less than 2 years diagnosis – $2^{nd}$ line $Vs.$ O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis² | XX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $1^{st}$ line Vs. O.B. – 2 years or more diagnosis – $1^{st}$ line <sup>3</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more diagnosis – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |


Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gr | oup | 2 <sup>nd</sup> g | roup | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** | Total no-missing* | Time to first intensification** | |
| | n | Median(Q1,Q3) | √n ` | Median(Q1,Q3) | p-value*** |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Inflamatory – 1 <sup>st</sup> line <sup>3</sup> | xx | xx.x (xx.x, xx.x) | ille xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory – 2 <sup>nd</sup> line Vs. O.B. – Inflamatory – 2 <sup>nd</sup> line <sup>4</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating <sup>2</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Stricturing/Penetrating $-$ 1st line Vs. O.B. $-$ Stricturing/Penetrating $-$ 1st line | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| 3 | 4 | dille | | | |
| VDZ Stricturing/Penetrating $-2^{nd}$ line Vs. O.B. $-$ Stricturing/Penetrating $-2^{nd}$ | xx all | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| line <sup>4</sup> | 0, | | | | |
| uc | Use | | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 2 <sup>nd</sup> line Vs. VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ $-$ 2 years or more diagnosis $-$ 1 <sup>st</sup> line Vs. VDZ $-$ less than 2 years diagnosis $-$ 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** Median(Q1,Q3) | Total no-missing* | Time to first intensification** Median(Q1,Q3) | p-value*** |
| $\mbox{VDZ}-2$ years or more diagnosis – $2^{\mbox{\scriptsize nd}}$ line Vs. $\mbox{VDZ}-$ less than 2 years diagnosis – $2^{\mbox{\scriptsize nd}}$ line $^{1}$ | xx | xx.x (xx.x, xx.x) | o xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| O.B. – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| O.B. – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis – 2 <sup>nd</sup> line <sup>1</sup> | xx only | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | XXX | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| $\text{O.B.}-2$ years or more diagnosis – $1^{\text{st}}$ line Vs. O.B. – less than 2 years diagnosis $1^{\text{st}}\text{line}^1$ | cial | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| $O.B2$ years or more diagnosis $-2^{nd}$ line Vs. $O.B$ less than 2 years diagnosis $2^{nd}$ line <sup>1</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ Vs. O.B. <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| diagnosis 2 <sup>nd</sup> line <sup>1</sup> VDZ Vs. O.B. <sup>5</sup> VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> line <sup>6</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



Study : EVOLVE


Date: 17FEB2022

| | 1 <sup>st</sup> gı | roup | 2 <sup>nd</sup> g | | |
|---|---|---|---|---|---|
| | Total no-missing* | Time to first intensification** | Total no-missing* | Time to first intensification** | |
| | n | Median(Q1,Q3) | ⊳n ` | Median(Q1,Q3) | p-value*** |
| /DZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | ille xx | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| /DZ – Extensive colitis – 2 <sup>nd</sup> line Vs. O.B. – Extensive colitis – 2 <sup>nd</sup> line <sup>7</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| DZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | xx | XX.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| DZ – less than 2 years diagnosis – 1 <sup>st</sup> line Vs. O.B. – less than 2 years | xx O <sub>U</sub> | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| agnosis – 1 <sup>st</sup> line <sup>6</sup> | 150 | | | | |
| DZ – less than 2 years diagnosis – 2 <sup>nd</sup> line Vs. O.B. – less than 2 years | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| iagnosis – 2 <sup>nd</sup> line <sup>7</sup> | cial xx | | | | |
| DZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis <sup>5</sup> | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| DZ - 2 years or more diagnosis $-1^{st}$ line Vs. O.B. $-2$ years or more diagnosis | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | X.XXXX |
| 1 <sup>st</sup> line <sup>6</sup> | | | | | |
| DZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more | xx | xx.x (xx.x, xx.x) | xx | xx.x (xx.x, xx.x) | x.xxxx |
| iagnosis – 2 <sup>nd</sup> line <sup>7</sup> | | | | | |

<sup>\*</sup>Patients with correct data to calculate "time to first intensification".

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II


<sup>\*\*</sup>Estimated with Kaplan-Meier method

<sup>\*\*\*</sup>Estimated with LogRank test.



<sup>1</sup>Data without PS-IPTW.

<sup>2</sup>Data with PS-IPTW (CD).

<sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).

<sup>5</sup>Data with PS-IPTW (UC).

<sup>6</sup>Data with PS-IPTW (UC-1<sup>st</sup> line).

<sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



# 9.4.7 Clinical response

Table 4.7.1 Clinical response at 14 weeks

| | 1 <sup>st</sup> group | | 2 <sup>nd</sup> ¢ | group | | |
|---|---|---|---|---|---|---|
| | | Patients with | *0 | Patients with | | |
| | Total no-missing | clinical response | Total no-missing | clinical response | | |
| | n | n(%) | n | n(%) | OR (IC95%)* | p-value* |
| CD | | 200 | 34. | | | |
| VDZ – 1 <sup>st</sup> line Vs. VDZ – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal Vs. VDZ – Colonic/Ileocolonic¹ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – Intensification Vs. VDZ – Colonic/Ileocolonic – Intesification¹ | Mexx Cigil | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Ileal – No Intensification Vs. VDZ – Colonic/Ileocolonic – No Intesification <sup>1</sup> | )Kx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis Vs. VDZ – less than 2 years diagnosis <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 years or more diagnosis – 1 <sup>st</sup> line Vs. VDZ – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| BIOCLEVER |
|-----------|

Study : EVOLVE


Date: 17FEB2022

| 1 <sup>st</sup> group | 2 <sup>nd</sup> group |
|-----------------------|-----------------------|
| Patients with | Patients with |

| | Total no-missing | clinical response | Total no-missing | clinical response | | |
|---|---|---|---|---|---|---|
| | n | n(%) | n ve | n(%) | OR (IC95%)* | p-value* |
| VDZ - 2 years or more diagnosis - $2^{nd}$ line Vs. VDZ - less than 2 years diagnosis - $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | xO' | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. VDZ – Stricturing/Penetrating <sup>1</sup> | xx | xx ( xx.x%) | JIDIE XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-Inflamatory-1^{st}\ line\ Vs.\ VDZ-Stricturing/Penetrating-1^{st}\ line^1$ | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| $VDZ$ – Inflamatory – $2^{nd}$ line $Vs.$ $VDZ$ – Stricturing/Penetrating – $2^{nd}$ line <sup>1</sup> | xx | xx (-xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal Vs. O.B. – Colonic/Ileocolonic <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic – 1 <sup>st</sup> line <sup>1</sup> | xx x | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic – 2 <sup>nd</sup> line <sup>1</sup> | ollili xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| O.B. – Ileal – Intensification Vs. O.B. – Colonic/Ileocolonic – Intesification <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Ileal – No Intensification Vs. O.B. – Colonic/Ileocolonic – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 2 years or more diagnosis Vs. O.B. – less than 2 years diagnosis <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II


O.B. – Inflamatory – 1<sup>st</sup> line Vs. O.B. – Stricturing/Penetrating – 1<sup>st</sup> line<sup>1</sup>

O.B. – Inflamatory – 2<sup>nd</sup> line Vs. O.B. – Stricturing/Penetrating – 2<sup>nd</sup>



#### STATISTICAL ANALYSIS PLAN

1<sup>st</sup> group

Study: EVOLVE


Date: 17FEB2022

X.XXXX

X.XXXX

| | | Patients with | | Patients with | | |
|---|---|---|---|---|---|---|
| | Total no-missing | clinical response | Total no-missing | clinical response | | |
| | n | n(%) | n Ne | n(%) | OR (IC95%)* | p-value* |
| O.B. $-2$ years or more diagnosis $-1$ <sup>st</sup> line Vs. O.B. $-$ less than 2 years diagnosis $1$ <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx <sub>O</sub> | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-2^{nd}$ line Vs. O.B. $-$ less than 2 years diagnosis $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | Jilije xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Inflamatory Vs. O.B. – Stricturing/Penetrating <sup>1</sup> | XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

xx ( xx.x%)

xx ( xx.x%)

xx.x (xx.x, xx.x)

xx.x (xx.x, xx.x)

| line <sup>1</sup> | . 2 | | | | | |
|---|---|---|---|---|---|---|
| VDZ Vs. O.B. <sup>2</sup> | e xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>4</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – Colonic/Ileocolonic Vs. O.B. – Colonic/Ileocolonic <sup>2</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxx |
| VDZ – Colonic/Ileocolonic – 1 <sup>st</sup> line Vs. O.B. – Colonic/Ileocolonic 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| inte | | | | | | |
| VDZ – Colonic/Ileocolonic – 2 <sup>nd</sup> line Vs. O.B. – Colonic/Ileocolonic 2 <sup>nd</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

line4

| BIOCLE! | ver |
|---------|-----|

Study : EVOLVE


Date: 17FEB2022

| 1 <sup>st</sup> gı | roup | 2 <sup>nd</sup> group |
|--------------------|-------------------|------------------------------------|
| | Patients with | Patients with |
| Total no-missing | clinical response | Total no-missing clinical response |

| | i otai no-missing | ciinicai response | lotal no-missing | ilnicai response | | |
|---|---|---|---|---|---|---|
| | n | n(%) | n (e) | n(%) | OR (IC95%)* | p-value* |
| VDZ – Ileal Vs. O.B. – Ileal² | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 1 <sup>st</sup> line Vs. O.B. – Ileal – 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | ×x xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Ileal – 2 <sup>nd</sup> line Vs. O.B. – Ileal – 2 <sup>nd</sup> line <sup>4</sup> | XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis² | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $1^{st}$ line Vs. O.B. – less than 2 years diagnosis – $1^{st}$ line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>4</sup> | w xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis² | OMMEXX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – $1^{st}$ line Vs. O.B. – 2 years or more diagnosis – $1^{st}$ line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more diagnosis – 2 <sup>nd</sup> line <sup>4</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Inflamatory Vs. O.B. – Inflamatory <sup>2</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

| | <i>Q</i> <sub>1</sub> |
|----------|-----------------------|
| | Study: EVOLVE |
| BIWLEVER | Date : 17FEB2022 |

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gro | oup Ole | | |
|---|---|---|---|---|---|---|
| | | Patients with | | Patients with | | |
| | Total no-missing | clinical response | Total no-missing | clinical response | | |
| | n | n(%) | n 🚫 | n(%) | OR (IC95%)* | p-value* |
| VDZ – Inflamatory – 1 <sup>st</sup> line Vs. O.B. – Inflamatory – 1 <sup>st</sup> line <sup>3</sup> | xx | xx ( xx.x%) | XX.O | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $\label{eq:VDZ-Inflamatory-2nd line Vs. O.BInflamatory-2^{nd line} \ ^4$ | XX | xx ( xx.x%) | XX XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating Vs. O.B. – Stricturing/Penetrating <sup>2</sup> | xx | xx ( xx.x%) | XX XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Stricturing/Penetrating – 1 <sup>st</sup> line Vs. O.B. – Stricturing/Penetrating | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| - 1 <sup>st</sup> line <sup>3</sup> | | KIL | | | | |
| VDZ Stricturing/Penetrating $-2^{nd}$ line Vs. O.B. $-$ Stricturing/Penetrating | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| – 2 <sup>nd</sup> line <sup>4</sup> | 19 | | | | | |
| UC | xx cial Us | | | | | |
| $VDZ - 1^{st}$ line $Vs. VDZ - 2^{nd}$ line <sup>1</sup> | exx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis Vs. VDZ – Proctitis/Left colitis <sup>1</sup> | July xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. VDZ – Proctitis/Left colitis – 1 <sup>st</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| line <sup>1</sup> | | | | | | |
| $VDZ$ – Extensive colitis – $2^{nd}$ line $Vs$ . $VDZ$ – $Proctitis/Left$ colitis – $2^{nd}$ | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| line <sup>1</sup> | | | | | | |
| VDZ – Extensive colitis – Intensification Vs. VDZ – Proctitis/Left colitis | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| - Intesification <sup>1</sup> | | | | | | |



1<sup>st</sup> group

Study : EVOLVE


Date: 17FEB2022

| | Total no-missing | Patients with clinical response | Total no-missing | Patients with | |
|---|---|---|---|---|---|
| | n | n(%) | n (© | n(%) | OR (IC95%)* |
| eft | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x |

2<sup>nd</sup> group

| | n | n(%) | n ve | n(%) | OR (IC95%)* | p-value* |
|---|---|---|---|---|---|---|
| VDZ – Extensive colitis – No Intensification Vs. VDZ – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. VDZ - less than 2 years diagnosis <sup>1</sup> | xx | xx ( xx.x%) | , ole xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ-2 years or more diagnosis – 1 <sup>st</sup> line Vs. $VDZ$ – less than 2 years diagnosis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $VDZ-2$ years or more diagnosis $-2^{nd}$ line $Vs.\ VDZ-less$ than 2 years diagnosis $-2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – 1 <sup>st</sup> line Vs. O.B. – 2 <sup>nd</sup> line <sup>1</sup> | xeigh | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis Vs. O.B. – Proctitis/Left colitis <sup>1</sup> | XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis – 1 <sup>st</sup> line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – $2^{nd}$ line Vs. O.B. – Proctitis/Left colitis – $2^{nd}$ line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. – Extensive colitis – Intensification Vs. O.B. – Proctitis/Left colitis – Intesification¹ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |



1<sup>st</sup> group

Study : EVOLVE


Date: 17FEB2022

| | Patients with | Pati | ents with | |
|---|---|---|---|---|
| Total no-missing | clinical response | Total no-missing clinical | al respons | e |
| n | n(%) | n ve | n(%) | OR (IC9 |

2<sup>nd</sup> group

| | Total no-missing | clinical response | Total no-missing | linical response | | |
|---|---|---|---|---|---|---|
| | n | n(%) | n we' | n(%) | OR (IC95%)* | p-value* |
| O.B. – Extensive colitis – No Intensification Vs. O.B. – Proctitis/Left colitis – No Intesification <sup>1</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $O.B 2$ years or more diagnosis Vs. $O.B less$ than 2 years diagnosis $^1$ | xx | xx ( xx.x%) | Jiloje xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-1^{st}$ line Vs. O.B. $-$ less than 2 years diagnosis $1^{st}$ line <sup>1</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| O.B. $-2$ years or more diagnosis $-2^{\text{nd}}$ line Vs. O.B. $-$ less than 2 years diagnosis $2^{\text{nd}}$ line <sup>1</sup> | xx S | xx ( xx.x%) | хх | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ Vs. O.B. <sup>5</sup> | xxidi | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. O.B. 1 <sup>st</sup> line <sup>6</sup> | Wexx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. O.B. 2 <sup>nd</sup> line <sup>7</sup> | offic xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – Proctitis/Left colitis Vs. O.B. – Proctitis/Left colitis <sup>5</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Proctitis/Left colitis – 1 <sup>st</sup> line Vs. O.B. – Proctitis/Left colitis 1 <sup>st</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| line <sup>6</sup> VDZ – Proctitis/Left colitis – 2 <sup>nd</sup> line Vs. O.B. – Proctitis/Left colitis 2 <sup>nd</sup> line <sup>7</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |

| | $Q_1$ |
|----------|------------------|
| | Study : EVOLVE |
| Bl@Lever | Date : 17FEB2022 |

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> gr | oup No | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Patients with clinical response | Total no-missing | Patients with | | |
| | n | n(%) | n © | n(%) | OR (IC95%)* | p-value* |
| VDZ – Extensive colitis Vs. O.B. – Extensive colitis <sup>5</sup> | xx | xx ( xx.x%) | xxO | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – Extensive colitis – 1 <sup>st</sup> line Vs. O.B. – Extensive colitis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | XX XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| $\label{eq:VDZ-Extensive} VDZ-Extensive \ colitis-2^{nd} \ line \ Vs. \ O.BExtensive \ colitis-2^{nd} \ line^7$ | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis Vs. O.B. – less than 2 years diagnosis <sup>5</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $1^{st}$ line Vs. O.B. – less than 2 years diagnosis – $1^{st}$ line <sup>6</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – less than 2 years diagnosis – $2^{nd}$ line Vs. O.B. – less than 2 years diagnosis – $2^{nd}$ line <sup>7</sup> | Musicial D. | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis Vs. O.B. – 2 years or more diagnosis <sup>5</sup> | ominexx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 1 <sup>st</sup> line Vs. O.B. – 2 years or more diagnosis – 1 <sup>st</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ - 2 years or more diagnosis – 2 <sup>nd</sup> line Vs. O.B. – 2 years or more diagnosis – 2 <sup>nd</sup> line <sup>7</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |

<sup>\*</sup>Estimated with a logistic regression.

¹Data without PS-IPTW.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | Study : EVOLVE |
|----------|------------------|
| BIWLEVEI | Date : 17FEB2022 |

0.

<sup>2</sup>Data with PS-IPTW (CD).

<sup>3</sup>Data with PS-IPTW (CD-1<sup>st</sup> line).

<sup>4</sup>Data with PS-IPTW (CD-2<sup>nd</sup> line).

<sup>5</sup>Data with PS-IPTW (UC).

<sup>6</sup>Data with PS-IPTW (UC-1<sup>st</sup> line).

<sup>7</sup>Data with PS-IPTW (UC-2<sup>nd</sup> line).

Table 4.7.2 Clinical response at 52 weeks

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II

| | | , 1/5° | Study : EVOLVE |
|----------|---------------------------|--------|------------------|
| | STATISTICAL ANALYSIS PLAN | Ó | Version : 6.0 |
| BIWLEVEI | | ins | Date : 17FEB2022 |

Table 4.7.3 CD patients with VDZ – Clinical response at 52 weeks Logistic regression-model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| odel | and Subject to | XX XX | |
| ne treatment | **0 | <b>~</b> | x.xxxx |
| pe of diagnosis | Nie Ct | | x.xxxx |
| ease duration | SILL | | x.xxxx |
| pe of disease behaviour at diagnosis | ano | | x.xxxx |
| eraction Line treatment and Type of diagnosis | 4 | | x.xxxx |
| eraction Line treatment and Disease duration eraction Line treatment and Type of disease behaviour at diagnosis eraction Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Line treatment, Type of diagnosis and Disease duration | | | x.xxxx |
| eraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |
| eraction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | Study : EVOLVE |
|----------|------------------|
| BIWLEVEI | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

Table 4.7.4 CD patients with VDZ – Clinical response at 52 weeks Logistic regression model (estimated OR)

| | *** | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | 2nd line Vs. 1st line Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Se | |
| 2 <sup>nd</sup> line | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Ileal Vs. Colonic/leocolonic | xx.x (xx.x, xx.x) |
| | alle | |

Note: Only significant variables and/or interactions (Table 4.6.5) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | Study: EVOLVE |
|----------|------------------|
| Bl@Lever | Date : 17FEB2022 |

Table 4.7.5 UC patients with VDZ - Clinical response at 52 weeks Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | xx xx | |
| ine treatment | | **0 | x.xxxx |
| Type of diagnosis | | | x.xxxx |
| Disease duration | Subje | | x.xxxx |
| nteraction Line treatment and Type of diagnosis | allo | | x.xxxx |
| nteraction Line treatment and Disease duration | Kling | | x.xxxx |
| nteraction Type of diagnosis and Disease duration | | | x.xxxx |
| nteraction Line treatment, Type of diagnosis and Disease duration | 7/2 | | x.xxxx |

| | | | Study : EVOLVE |
|----------|---------------------------|----|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | MS | Date : 17FEB2022 |

Table 4.7.6 UC patients with VDZ - Clinical response at 52 weeks Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | SUDIE | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| | 81 | |

Note: Only significant variables and/or interactions (Table 4.6.7) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | , 150 | Study : EVOLVE |
|----------|-------|------------------|
| BIWLEVER | MS | Date : 17FEB2022 |

Table 4.7.7 CD patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| odel | xx | xx xx | |
| ne treatment | and sulpiection | <u>~</u> | x.xxxx |
| e of diagnosis | Niec, | | x.xxxx |
| ease duration | Sull' | | x.xxxx |
| e of disease behaviour at diagnosis | 2100 | | x.xxxx |
| raction Line treatment and Type of diagnosis | | | x.xxxx |
| eraction Line treatment and Disease duration eraction Line treatment and Type of disease behaviour at diagnosis eraction Type of diagnosis and Disease duration | | | x.xxxx |
| raction Line treatment and Type of disease behaviour at diagnosis | | | x.xxxx |
| raction Type of diagnosis and Disease duration | | | x.xxxx |
| raction Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxxx |
| raction Disease duration and Type of disease behaviour at diagnosis | | | x.xxx |
| eraction Line treatment, Type of diagnosis and Disease duration | | | x.xxx |
| eraction Line treatment, Type of diagnosis and Type of disease behaviour at diagnosis | | | x.xxx |
| raction Line treatment, Disease duration and Type of disease behaviour at diagnosis | | | x.xxx |
| raction Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | | Study: EVOLVE |
|-------------|---------------------------|------------------|
| DISOLON (OK | STATISTICAL ANALYSIS PLAN | Version : 6.0 |
| Bl@Lever | | Date : 17FEB2022 |

| | n | Missing | p-value |
|---|---|---|---|
| Interaction Line treatment, Type of diagnosis, Disease duration and Type of disease behaviour at diagnosis | | | x.xxxx |

Table 4.7.8 CD patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (estimated OR)

| | | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | 2nd line Vs. 1st line Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Type of disease behaviour at diagnosis | Inflammatory Vs. Stricturing / Penetrating | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Se | |
| 2 <sup>nd</sup> line | lleal Vs. Colonic/lleocolonic | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Ileal Vs. Colonic/Ileocolonic | xx.x (xx.x, xx.x) |
| | alle | |

Note: Only significant variables and/or interactions (Table 4.6.5) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | $\mathcal{O}_1$ |
|----------|------------------|
| | Study : EVOLVE |
| BIWLEVER | Date : 17FEB2022 |

Table 4.7.9 UC patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (p-values)

| | n | Missing | p-value |
|---|---|---|---|
| Model | xx | **/© xx | |
| Line treatment | | ,00 | x.xxxx |
| Type of diagnosis | i,e <sup>C</sup> | | x.xxxx |
| Disease duration | Subjec | | x.xxx |
| Interaction Line treatment and Type of diagnosis | and | | x.xxxx |
| Interaction Line treatment and Disease duration | KING | | x.xxx |
| Interaction Type of diagnosis and Disease duration | °⊗<br>O, | | x.xxxx |
| Interaction Line treatment, Type of diagnosis and Disease duration | 1/2 | | x.xxxx |

| | | | Study : EVOLVE |
|----------|---------------------------|----|------------------|
| | STATISTICAL ANALYSIS PLAN | Ö | Version : 6.0 |
| BIWLEVER | | MS | Date : 17FEB2022 |

Table 4.7.10 UC patients with Other Biologic – Clinical response at 52 weeks Logistic regression model (estimated OR)

| | , | OR (CI 95%) |
|---|---|---|
| Line Treatment | 2nd line Vs. 1st line | xx.x (xx.x, xx.x) |
| Type of diagnosis | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| Line Treatment | 2 years or more Vs. less than 2 years | xx.x (xx.x, xx.x) |
| Interaction Line treatment and Type of diagnosis | Subje | |
| 2 <sup>nd</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| 1 <sup>st</sup> line | Extensive colitis Vs. Proctitis/Left colitis | xx.x (xx.x, xx.x) |
| | 8) | |

Note: Only significant variables and/or interactions (Table 4.6.7) will be included in this table.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# 9.4.8 Clinical remission

# Table 4.8.1 Clinical remission at 14 weeks

Table 4.8.2 Clinical remission at 52 weeks

Table 4.8.3 CD patients with VDZ – Clinical remission at 52 weeks Logistic regression model (p-values)

Table 4.8.4 CD patients with VDZ - Clinical remission at 52 weeks Logistic regression model (estimated OR)

Table 4.8.5 UC patients with VDZ - Clinical remission at 52 weeks Logistic regression model (p-values)

Table 4.8.6 UC patients with VDZ - Clinical remission at 52 weeks Logistic regression model (estimated OR)

Table 4.8.7 CD patients with Other Biologic Clinical remission at 52 weeks Logistic regression model (p-values)

Table 4.8.8 CD patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (estimated OR)

Table 4.8.9 UC patients with Other Biologic – Clinical remission at 52 weeks Logistic regression model (p-values)

Table 4.8.10UC patients with Other Biologic - Clinical remission at 52 weeks Logistic regression model (estimated OR)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# 9.4.9 Endoscopic response at 52 weeks

# Table 4.9.1 Endoscopic response at 52 weeks

Table 4.9.2 CD patients with VDZ - Endoscopic response at 52 weeks Logistic regression model (p-values)

Table 4.9.3 CD patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (estimated OR)

Table 4.9.4 UC patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (p-values)

Table 4.9.5 UC patients with VDZ – Endoscopic response at 52 weeks Logistic regression model (estimated OR)

Table 4.9.6 CD patients with Other Biologic – Endoscopic response at 52 weeks Logistic regression model (p-values)

Table 4.9.7 CD patients with Other Biologic – Endoscopic response at 52 weeks Logistic regression model (estimated OR)

Table 4.9.8 UC patients with Other Biologic - Endoscopic response at 52 weeks Logistic regression model (p-values)

Table 4.9.9 UC patients with Other Biologic – Endoscopic response at 52 weeks Logistic regression model (estimated OR)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# 9.4.10 Endoscopic remission at 52 weeks

Table 4.10.1Endoscopic remission at 52 week

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# 9.4.11 Biochemical remission based on CRP

Table 4.11.1Biochemical remission based on CRP at 14 weeks

Table 4.11.2Biochemical remission based on CRP at 52 weeks

9.4.12 Biochemical remission based on fecal calprotectin

Table 4.12.1Biochemical remission based on fecal calprotectin at 14 weeks

Table 4.12.2Biochemical remission based on fecal calprotectin at 52 weeks

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



# 9.5 Secondary objectives

9.5.1 Describe the real world clinical effectiveness of VDZ vs. other biologics at least 12 months post-treatment initiation (in a subgroup of patients with adequate follow-up available)

Included in section 9.4.

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II



Study: EVOLVE

Date: 17FEB2022


# 9.5.2 Quantify healthcare resource utilization including the rates of healthcare erns of Use professional (HCP) and emergency department (ED) visits, hospitalizations and Inflammatory Bowel Disease (IBD) related surgical procedures

Table 5.2.1 Health resource utilization - CD with VDZ patients

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Any visit? | | .0 | PA |
| Total no-missing | n | xx voluge | XX |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx:x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n 150 | xx | xx |
| | i a | | |
| Yes 1 2 Missing /isit of:* Total no-missing Emergency doctor 1 2 Specialist | Reko | | |
| Total no-missing | offin n | xx | xx |
| Emergency doctor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 695. | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Specialist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Surgery | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index<br>date and index date<br>(n=xx) | 12 months Post-<br>Index date<br>(n=xx) |
|---|---|---|---|
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Diagnostic test | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission | n (%) | xx ( xx.x%) | XX ( XX.X%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx, x%) | xx ( xx.x%) |
| Hospital admission (with | n (%) out n (%) n (%) n (%) n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | nicita | xx | xx |
| Visit with professional:* | Stull | | |
| Total no-missing Internist 1 2 General Practitioner | n | xx | XX |
| Internist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| General Practitioner | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Visit with surgery:* | | | |
| Total no-missing | n | XX | xx < |
| Resection | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Resection with ostomy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx,x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | OUB | |
| | SO | | |
| Visit with diagnostic test:* | | | |
| Total no-missing | n (%) n (%) | xx | xx |
| Endoscopy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Endoscopy 1 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 401 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Kor, | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| MRI MRI POT MOTO | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 3/Les | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Any visit with hospitalization? | | | |
| Total no-missing | n | xx | xx |




Date : 17FEB2022

XX

12 months Post-12 months pre -Index date and index date Index date (n=xx)(n=xx)No n (%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) Yes n (%) 1 n (%) xx ( xx.x%) 2 n (%) xx ( xx.x%) xx ( xx.x%) n (%) Missing n Number of hospitalization days  $n^1$ XX Mean (SD) xx.x (xx.x) Median (Q1, Q3) xx.x (xx.x, xx.x) Min, Max XX, XX

Table 5.2.2 Health resource utilization related to the pathology – CD with VDZ patients

Missing

| | Collings | 12 months pre -Index<br>date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Any visit? | ) | | |
| Total no-missing | n | xx | xx |
| Total no-missing No Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 0 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

Visit of:\*

<sup>&</sup>lt;sup>1</sup>Number of visits.



Study : EVOLVE

Date : 17FEB2022


| | | 12 months pre -Index<br>date and index date<br>(n=xx) | 12 months Post-<br>Index date<br>(n=xx) |
|---|---|---|---|
| Total no-missing | n | xx | xx |
| Emergency doctor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Specialist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx.(*xx,x%) | xx ( xx.x%) |
| Surgery | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) n (%) n (%) n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Diagnostic test | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | nr(%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 Hospital admission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission (without | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission (without | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| surgery) | | | |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |



Total no-missing

## STATISTICAL ANALYSIS PLAN

Study : EVOLVE


Date : 17FEB2022

12 months pre -Index 12 months Postdate and index date Index date Terms of Use (n=xx) (n=xx)Visit with professional:\* Total no-missing n XXInternist n (%) xx ( xx.x%) 1 n (%) xx (xx.x%) 2 n (%) xx (xx.x%) xx ( xx.x%) xx ( xx.x%) n (%) **General Practitioner** xx ( xx.x%) xx ( xx.x%) n (%) For Monrooming rolal Use Only and some oster n (%) xx ( xx.x%) 2 xx ( xx.x%) xx (xx.x%) Visit with surgery:\* Total no-missing XXXXResection xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) 2 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) Resection with ostomy xx ( xx.x%) n (%) xx ( xx.x%) n (%) xx ( xx.x%) xx ( xx.x%) n (%) xx ( xx.x%) xx ( xx.x%) n (%) xx ( xx.x%) xx ( xx.x%) Visit with diagnostic test:\*

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

ХX

ХX

n



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Endoscopy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| MRI | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | <i>GUDIPE</i> | |
| Any visit with hospitalization? | | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | |
| Total no-missing | n Or | xx | XX |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | | xx ( xx.x%) | xx ( xx.x%) |
| 2 Missing | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | XX |
| 401 | | | |
| Number of hospitalization days | n¹ | xx | XX |
| 1 ste | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Missing Number of hospitalization days | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| | Missing | XX | xx |

<sup>&</sup>lt;sup>1</sup>Number of visits.



Study: EVOLVE

Date: 17FEB2022


Table 5.2.3 Health resource utilization - CD patients with other biologic

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Any visit? | | | |
| Total no-missing | n | xx | xx © |
| No | n (%) | xx ( xx.x%) | xx ( xx x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx x%) | xx ( xx.x%) |
| Missing | n | SUXX | xx |
| | | and | |
| Visit of:* | | xx (xx.x%) | |
| Total no-missing | n | xx | xx |
| Emergency doctor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 2 Specialist 1 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Specialist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 2 Surgery | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Leoc | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Surgery | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Diagnostic test | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index<br>date and index date<br>(n=xx) | 12 months Post-<br>Index date<br>(n=xx) |
|---|---|---|---|
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | XX ( XX.X%) |
| Hospital admission (wit | thout n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | Cxx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n ( | OUT XX | xx |
| Visit with professional:* | n (%) | | |
| Total no-missing | n (C) | xx | xx |
| Internist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 General Practitioner 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| General Practitioner | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Visit with surgery:* | | | |
| Total no-missing | n | xx | xx |



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Resection | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Resection with ostomy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | | 1018 | |
| | | 50 | |
| Visit with diagnostic test:* | | 1 Sille | |
| Total no-missing | n | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx |
| Endoscopy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | 4O, | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| MRI | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| MRI 1 2 MRI 1 2 And the day | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 99. | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| XXX | | | |
| O. | | | |
| Any visit with hospitalization? | | | |
| Total no-missing | n | xx | xx |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx < |
| | | | Slices Le |
| Number of hospitalization days | n¹ | xx | JICXX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |
| | Missing | XX | xx |

<sup>&</sup>lt;sup>1</sup>Number of visits.

Table 5.2.4 Health resource utilization related to the pathology – CD patients with other biologic

| | 150 | 12 months pre -Index | 12 months Post- |
|---|---|---|---|
| | | date and index date | Index date |
| | Cio | (n=xx) | (n=xx) |
| Any visit? | n (%) n (%) n (%) n (%) n (%) n (%) n (%) | | |
| Total no-missing | CO n | xx | XX |
| No Wor | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 160 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| <u> </u> | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| Visit of:* | | | |
| Total no-missing | n | xx | XX |
| Emergency doctor | n (%) | xx ( xx.x%) | xx ( xx.x%) |



Study : EVOLVE


Date: 17FEB2022

| 1 | (n=xx) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | (n=xx) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) |
|---|---|---|
| 2 | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| n (%) Specialist n (%) 1 n (%) 2 n (%) n (%) Surgery n (%) | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Specialist n (%) 1 n (%) 2 n (%) n (%) Surgery n (%) | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| 1 n (%) 2 n (%) n (%) Surgery n (%) | xx ( xx.x%)<br>xx ( xx.x%) | xx (xx.x%) |
| 2 n (%) n (%) Surgery n (%) | xx ( xx.x%) | .06, |
| n (%) Surgery n (%) | | xx ( xx.x%) |
| Surgery n (%) | xx ( xx.x%) | <b>*</b> |
| | <b>,</b> ,, | xx ( xx.x%) |
| 1 n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx,x%) | xx ( xx.x%) |
| 2 n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Diagnostic test n (%) | OKIIS xx ( xx.x%) | xx ( xx.x%) |
| 1 n (%) | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%) |
| 2 n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n(%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital admission 1 | xx ( xx.x%) | xx ( xx.x%) |
| 2 n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Hospital Admission (without n (%) | xx ( xx.x%) | xx ( xx.x%) |
| surgery | | |
| n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 n (%) | xx ( xx.x%) | xx ( xx.x%) |
| n (%) | ( | xx ( xx.x%) |
| Missing n | xx ( xx.x%) | , |

Visit with professional:\*



Study : EVOLVE


Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Post-<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| Total no-missing | n | xx | XX |
| Internist | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| General Practitioner | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx (*xx,x%) | xx ( xx.x%) |
| | | 250 | |
| | | and | |
| Visit with surgery:* | | xx (xx.x%) xx xx (xx.x%) | |
| Total no-missing | n S | xx | xx |
| Resection | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Resection with ostomy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 Resection with ostomy 1 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 80. | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| X OX | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Visit with diagnostic test:* | | | |
| Total no-missing | n | xx | xx |
| Endoscopy | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |




Date: 17FEB2022

| | | 12 months pre -Index date and index date | 12 months Pos<br>Index date |
|---|---|---|---|
| | | (n=xx) | (n=xx) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| MRI | n (%) | xx ( xx.x%) | xx ( xx.x%)/ |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | XX ( xx.x%) |
| | | ille | |
| | | xx (xx.x%) xx (xx.x%) | |
| Any visit with hospitalization? | | ibiles | |
| Total no-missing | n n (%) n (%) n (%) n (%) | xx | xx |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 | n (%)<br>n (%)<br>n | xx ( xx.x%) | xx ( xx.x%) |
| | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |
| | , | | |
| Number of hospitalization days | n¹ | xx | xx |
| 40 | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| 890. | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x |
| Number of hospitalization days 1 Number of visits. | Min, Max | xx, xx | xx, xx |
| S. T. | Missing | xx | XX |



Journe utilization – UC patients with VDZ

Lation related to the pathology – UC patients with VDZ

Jealth resource utilization – CD patients with other biologic

A resource utilization related to the pathology – UC patients with other biologic

A resource utilization related to the pathology – UC patients with other biologic

A propagation of the pathology – UC patients with other biologic

A pathology – UC patients with other biologic

A patients with VDZ

A patients with vDZ

A patients with vDZ

A patients with vDZ

A patients with other biologic

A patients with other biologic

A patients with other biologic

A patients with vDZ

A p

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




# Properly of Takeda: For Mon. Commercial Use Only and Subject to the Applicable Terms of Use



Study: EVOLVE

Date: 17FEB2022


9.5.4 Describe treatment patterns, clinical effectiveness and safety events for Table 5.4.1 Patients who discontinue index treatment in the VDZ cohort and initiate a second-line biologic within 6 months post-index treatment discontinuation at least the induction phase of the subsequent biologic regimen for

| Patients with treatment discontinuation Total no-missing n xx total results with treatment discontinuation Yes n (%) xx (xx x%) No n (%) xx (xx x%) Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx x%) No n (%) xx (xx x%) Missing n xx ¹Patients with treatment discontinuation. | VDZ (UC<br>(n=xx) |
|---|---|
| Patients with treatment discontinuation Total no-missing n xx Yes n (%) xx (xx/x%) No n (%) xx (xx/x%) Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) No xx (xx.x%) Missing n xx | (n=xx) |
| Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) No x (xx.x%) No x (xx.x%) | ZP ( 2) |
| Yes n (%) xx (xxxx%) No n (%) xx (xxxx%) Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xxxx%) No n (%) xx (xxxx%) Missing n xx | <b>y</b> |
| No n (%) xx (xx.x%) Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | xx |
| Missing n xx Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | xx ( xx.x% |
| Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | xx ( xx.x% |
| Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | xx |
| Patients who initiate a new-line biologic within 6 months post-index treatment discontinuation¹ Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | |
| Total no-missing n xx Yes n (%) xx (xx.x%) No n (%) xx (xx.x%) Missing n xx | |
| No n (%) xx ( xx.x%) Missing n xx | |
| No n (%) xx ( xx.x%) Missing n xx | xx |
| No n (%) xx ( xx.x%) Missing n xx | xx ( xx.x% |
| 70 | xx ( xx.x% |
| <sup>1</sup> Patients with treatment discontinuation. | xx |
| K Lakedai. Fo. | |
| K Lakeda. | |
| of Steel | |
| ,0 | |



Study : EVOLVE

Date: 17FEB2022


# **Table 5.4.1 New treatment**

| | l able 5.4.1 | New treatment | |
|---|---|---|---|
| | | VDZ with new treatment within 6 months post-index treatment discontinuation (CD) | VDZ with new treatment within 6 months post-index treatment discontinuation (UC) |
| | | (n=xx) | (n=xx) |
| Time from index date to new treatmet (months) | ent n | xx | COPIIC® S |
| | Mean (SD) | xx.x (xx.x) | ×x.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | XX, XX |
| | Missing | XX.X (XX.X, XX.X) XX, XX XX XX | xx |
| Time from treatment discontinuation to ne | ew n | Sille XX | xx |
| treatment (months) | OUB | | |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (Q1, Q3) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Min, Max | xx, xx | xx, xx |
| Oncomin | Missing | xx | xx |
| Patients with treatment discontinuation | | | |
| Total no-missing | n | xx | xx |
| Golimumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Ceertolizumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Infliximab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Ustekinumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Tofacitinib | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Adalimumab | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n | xx | xx |

<sup>&</sup>lt;sup>1</sup>Patients with treatment discontinuation



Study : EVOLVE

Date: 17FEB2022


Table 5.4.2 Posology (mg) by treatment

| | n | Media<br>(Desv. estándar) | Mediana<br>(Q1, Q3) | Min, Max | Missing |
|---|---|---|---|---|---|
| CD | | | | | |
| Golimumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Ceertolizumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | xx © |
| Infliximab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | Olexx |
| Ustekinumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | xx |
| Tofacitinib | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Adalimumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| UC | | | Č. | Q | |
| Golimumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Ceertolizumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Infliximab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Ustekinumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | XX, XX | XX |
| Tofacitinib | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | xx, xx | XX |
| Adalimumab | xx | xx.x (xx.x) | xx.x (xx.x, xx.x) | XX, XX | XX |
| of akedai. | xx Hon-C | omine. | | | |




Date: 17FEB2022

# Table 5.4.1 New treatment - Response and remission 14 weeks

| - | | | |
|---|---|---|---|
| | | VDZ with new treatment within 6 months post-index treatment discontinuation (CD) | VDZ with new treatment within 6 months post-index treatment discontinuation (UC) |
| Response at 14 weeks | | (n=xx) | (n=xx) |
| Total no-missing | n | XX | oplice xx |
| Yes | | | XX ( XX.X%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n (70) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X70) |
| Remission at 14 weeks | | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | |
| Total no-missing | n H | xx | xx |
| Yes | | xx ( xx.x%) | xx ( xx.x%) |
| No | n (%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | n n | xx | xx |
| Missing Korkedai. For Work. Company of Lakedai. | | | |




Date: 17FEB2022

## Table 5.4.2 New treatment - Adverse Events

VDZ with new treatment within 6 months post-index treatment discontinuation (CD)

VDZ with new treatment within 6 months post-index treatment discontinuation (UC)

(n=xx)(n=xx)

| | Total no-missing | Patients with any AE | Total no-missing | Patients with any AE |
|---|---|---|---|---|
| | n | n(%) | n | n(%) |
| Adverse event | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse | xx | xx ( xx.x%) | xx | <b>※</b> x ( xx.x%) |
| event r | | | | SPA |
| Adverse event | xx | xx ( xx.x%) | xx xx xx xx xx xx | xx ( xx.x%) |
| related with | | | a XXO | |
| treatment | | | iece | |
| Serious Adverse | xx | xx ( xx.x%) | SILO XX | xx ( xx.x%) |
| event related with | | 50 | > | |
| treatment | | 31, | | |
| Infections, serious | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| infections and | | 01 | | |
| malignancies | | 72 | | |
| Note: Adverse Ever | Nou-Country | | | |
| this | | | | |



| | Tabl | e 5.5.1 Adverse Events | No by | |
|---|---|---|---|---|
| | \ | /DZ | Other | Biologic |
| | Total no-missing | Patients with any AE | Total no-missing | Patients with any AE |
| | n | n(%) | n | n(%) |
| D | | 29.2 | | |
| dverse event | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| erious Adverse event r | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| dverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| erious Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| fections, serious infections and malignancies | xx dell | xx ( xx.x%) | xx | xx ( xx.x%) |
| D 1 <sup>st</sup> line | COMI | | | |
| dverse event | For Morkx | xx ( xx.x%) | xx | xx ( xx.x%) |
| erious Adverse event r | ×× ×× | xx ( xx.x%) | xx | xx ( xx.x%) |
| dverse event related with treatment | <b>₹</b> ○` xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| erious Adverse event related with treatment | × | xx ( xx.x%) | XX | xx ( xx.x%) |
| nfections, serious infections and malignancies | XX | xx ( xx.x%) | XX | xx ( xx.x%) |




Study : EVOLVE


Date: 17FEB2022

| | v | DZ | Other Biologic | |
|---|---|---|---|---|
| | Total no-missing | Total no-missing Patients with any AE | | Patients with any AE |
| | n | n(%) | DQ n | n(%) |
| CD 2 <sup>nd</sup> line | | | io ine xx | |
| Adverse event | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event r | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Infections, serious infections and malignancies | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| UC | | 150 | | |
| Adverse event | xx | xx ( xx.x%)<br>xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event r | xx cerc. | xx ( xx.x%) | xx | xx ( xx.x%) |
| Adverse event related with treatment | xx offile | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event related with treatment | ×C × | xx ( xx.x%) | xx | xx ( xx.x%) |
| Infections, serious infections and malignancies | * 40, xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| UC 1 <sup>st</sup> line | ₹0, | | | |
| Adverse event | Kot Mouxx<br>xx xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event r | xx | xx ( xx.x%) | xx | xx ( xx.x%) |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II




Study : EVOLVE


Date: 17FEB2022

| | , | /DZ | Other | Biologic |
|---|---|---|---|---|
| | Total no-missing | Patients with any AE | Total no-missing | Patients with any AE |
| | n | n(%) | p.P.n | n(%) |
| Adverse event related with treatment | xx | xx ( xx.x%) | **// <sub>©</sub> xx | xx ( xx.x%) |
| Serious Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Infections, serious infections and malignancies | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| UC 2 <sup>nd</sup> line | | 300 | | |
| Adverse event | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event r | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Serious Adverse event related with treatment | xx | xx ( xx.x%) | xx | xx ( xx.x%) |
| Infections, serious infections and malignancies | xx & | xx ( xx.x%) | xx | xx ( xx.x%) |

| | | Study: EVOLVE |
|-------------|---------------------------|------------------|
| DISOLON (OK | STATISTICAL ANALYSIS PLAN | Version : 6.0 |
| Bl@Lever | | Date : 17FEB2022 |

Table 5.5.2 Adverse event (incidence)

| | 1 <sup>st</sup> | group | 2 <sup>nd</sup> 9 | roup | | |
|---|---|---|---|---|---|---|
| | | Patients with any | *0 | Patients with any | | |
| | Total no-missin | g AE | Total no-missing | AE | | |
| | n | n(%) | (D) n | n(%) | OR (IC95%)* | p-value* |
| CD | | 6 | | | | |
| VDZ Vs. Other Biologic <sup>1</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 1 <sup>st</sup> line Vs. Other Biologic 1 <sup>st</sup> line <sup>2</sup> | xx | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 2 <sup>nd</sup> line Vs. Other Biologic 2 <sup>nd</sup> line <sup>3</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| UC | Mexicial s | | | | | |
| VDZ Vs. Other Biologic <sup>4</sup> | (XX | xx ( xx.x%) | XX | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |
| VDZ – 1 <sup>st</sup> line Vs. Other Biologic 1 <sup>st</sup> line <sup>5</sup> | CORPUT XX | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. Other Biologic 2 <sup>nd</sup> line <sup>6</sup> | xx | xx ( xx.x%) | xx | xx ( xx.x%) | xx.x (xx.x, xx.x) | X.XXXX |

<sup>\*</sup>Estimated with a logistic regression.


<sup>&</sup>lt;sup>1</sup>Data with PS-IPTW (CD); <sup>2</sup>Data with PS-IPTW (CD-1st line); <sup>3</sup>Data with PS-IPTW (CD-2nd line)

 $<sup>^4</sup>$ Data with PS-IPTW (UC);  $^5$ Data with PS-IPTW (UC-1st line);  $^6$ Data with PS-IPTW (UC-2nd line)



Table 5.5.3 Serious Adverse event (incidence)

Table 5.5.4 Related with treatmetn Adverse Event (incidence)

Table 5.5.5 Related with treatment Serious Adverse Event (incidence)

Table 5.5.6 Adverse event - Infections, serious infections and malignancies (incidence)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


| | Study : EVOLVE |
|----------|------------------|
| Bl@Lever | Date : 17FEB2022 |

Table 5.5.1 Adverse event (incidence rate)

| | 1 <sup>st</sup> g | roup | 2 <sup>nd</sup> g | roup | | |
|---|---|---|---|---|---|---|
| | Total no-missing | Nº AEs | Total no-missing | Nº AEs | | |
| | n | 100 patient/year | Ç'n | 100 patient/year | RR (IC95%)* | p-value* |
| CD | | C | JOIS | | | |
| VDZ Vs. Other Biologic <sup>1</sup> | xx | x.xx | xx | xx ( xx.x%) | X.XX | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. Other Biologic 1 <sup>st</sup> line <sup>1</sup> | xx | x.xx | xx | xx ( xx.x%) | X.XX | x.xxxx |
| $VDZ - 2^{nd}$ line Vs. Other Biologic $2^{nd}$ line <sup>2</sup> | xx | O x.xx | XX | xx ( xx.x%) | X.XX | x.xxxx |
| UC | , \\\circ\circ\circ\circ\circ\circ\circ\c | | | | | |
| VDZ Vs. Other Biologic <sup>3</sup> | XX. | X.XX | xx | xx ( xx.x%) | X.XX | x.xxxx |
| VDZ – 1 <sup>st</sup> line Vs. Other Biologic 1 <sup>st</sup> line <sup>3</sup> | all exx | x.xx | xx | xx ( xx.x%) | X.XX | x.xxxx |
| VDZ – 2 <sup>nd</sup> line Vs. Other Biologic 2 <sup>nd</sup> line <sup>4</sup> | COLUMN XX | X.XX | XX | xx ( xx.x%) | X.XX | X.XXXX |

<sup>\*</sup>Estimated with a Poisson regression including the following time.

Table 5.5.2 Serious Adverse event (incidence rate)


<sup>&</sup>lt;sup>1</sup>Data with PS-IPTW (CD); <sup>2</sup>Data with PS-IPTW (CD-1st line); <sup>3</sup>Data with PS-IPTW (CD-2nd line)

<sup>&</sup>lt;sup>4</sup>Data with PS-IPTW (UC); <sup>5</sup>Data with PS-IPTW (UC-1st line); <sup>6</sup>Data with PS-IPTW (UC-2nd line)



Table 5.5.3 Related with index date Adverse Event (incidence rate)

Table 5.5.4 Related with index date Serious Adverse Event (incidence rate)

Table 5.5.5 Adverse event - Infections, serious infections and malignancies (incidence rate)

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


Study: EVOLVE

STATISTICAL ANALYSIS PLAN


Date: 17FEB2022

# Table 5.5.6 Adverse Events I – CD patients with VDZ

| | | | | | | Table 5. | J.O AUVEI | Se Events 1 - | - OD patien | its with VD2 | -1100 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Resol | ved | | AE seriousness criteria assessment | | | | | | |
| | | | | | | | | Causality/Relationship to study drug | | | | | |
| | | | | | | | | | Hosp. or | , O. | Congenital | | |
| | Nº pat. | Ν° | | | | Duration | | Life- | prolong. | Disability/ | anomaly/birth | Important | |
| | (%) | ΑE | Yes | No | Unkn. | (days)* | Death | threating | Hosp. | incapacity | defect | medical event | None |
| <u>verall</u> | xx (xx.x) | xx | хх | xx | xx | x.x (x.x) | xx | XX | xxSU | XX | xx | xx | xx |
| OC 1 | xx (xx.x) | xx | xx | XX | XX | x.x (x.x) | xx | XX | Si xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | XX | xx | xx | xx | x.x (x.x) | XX | \S <sup>®</sup> x | XX | xx | xx | XX | xx |
| OC 2 | xx (xx.x) | XX | xx | xx | xx | x.x (x.x) | a Wich | xx | XX | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | XX | xx | xx | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | XX |
| PT 2 | xx (xx.x) | XX | xx | xx | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| | | | | | | , of Horrison | | | | | | | |
| | | | | | < | ,0, | | | | | | | |

<sup>\*</sup>Mean (Standard Deviation).

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II




Table 5.5.7 Adverse Events II - CD patients with VDZ

| | | | Related | to index drug | | Action taken with VDZ | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Nº pat.<br>(%) | N°<br>AE | Yes | No | Trt. Withdrawn | Dose reduced | Dose increased | Dose delayed | Dose not changed | Unknown | Not<br>applicable |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | xx | xx | xx c | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | Sign | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | XX | xx di | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | XX | xx off | XX | xx | xx | xx | xx |
| SOC 2 | xx (xx.x) | xx | xx | XX | xx | 19°xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | XX XX | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx Inher | xx | xx | xx | xx | xx | xx |
| | | | | | Colui | | | | | | |




Table 5.5.8 Adverse Events III – CD patients with VDZ

### Outcome

| | | | | | | D.K. | | |
|---|---|---|---|---|---|---|---|---|
| | Nº pat. (%) | Nº AE | Recovered | Recovering | Not recovered | Recovered with | Fatal | Unknown |
| | N pat. (76) | N AL | Recovered | Recovering | Not recovered | sequelae | | |
| Overall | xx (xx.x) | xx | xx | xx | xx | xx xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx si | XX | XX | xx |
| PT 1 | xx (xx.x) | xx | xx | XX | xx and | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | XX | - M.O. | xx | XX | xx |
| | | | | | 0, | | | |
| SOC 2 | xx (xx.x) | xx | xx | xx | US® XX | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx cic | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | W. W. W. C. | xx | xx | xx | xx |
| | | | | Coll. | | | | |

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.


Study: EVOLVE

STATISTICAL ANALYSIS PLAN


Date: 17FEB2022

# Table 5.5.9 Adverse Events I – CD patients with Other Biologic

| | | | | Resol | ved | | | | AE | seriousness c | riteria assessment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Са | usality/Relation | ship to study drug | | |
| | | | | | | | | | Hosp. or | *O | Congenital | | |
| | Nº pat. | Nº | | | | Duration | | Life- | prolong. | Disability/ | anomaly/birth | Important | |
| | (%) | ΑE | Yes | No | Unkn. | (days)* | Death | threating | Hosp. | incapacity | defect | medical event | None |
| Overall | xx (xx.x) | xx | xx | xx | XX | x.x (x.x) | xx | xx | xxS)), | XX | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | XX | XX | XX | x.x (x.x) | xx | xx | SLXX | xx | XX | xx | XX |
| PT 1 | xx (xx.x) | xx | XX | xx | xx | x.x (x.x) | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | XX | XX | XX | xx | x.x (x.x) | XX | Sex | XX | XX | xx | xx | xx |
| | | | | | | | :32 | | | | | | |
| SOC 2 | xx (xx.x) | XX | XX | XX | XX | x.x (x.x) | XXC. | xx | xx | xx | XX | xx | XX |
| PT 1 | xx (xx.x) | xx | xx | xx | XX | x.x (x.x) | ni xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | XX | xx | xx | x.x (x.x) | xx | xx | xx | xx | XX | xx | XX |

\*Mean (Standard Deviation).

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.




Table 5.5.10Adverse Events II - CD patients with Other Biologic

| | | | Related | to index drug | | Action taken with Other Biologic | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Nº pat.<br>(%) | N°<br>AE | Yes | No | Trt. Withdrawn | Dose reduced | Dose increased | Dose delayed | Dose not changed | Unknown | Not<br>applicable |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | xx | xx | xx. ect | xx | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | xx | S**018 | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | nd xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | хх | xx ofth | xx | xx | xx | xx | xx |
| SOC 2 | xx (xx.x) | xx | xx | xx | xx | 120xx | xx | xx | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx | xx (S) | xx | xx | xx | xx | xx | xx |
| | | | | | Colu | | | | | | |




Table 5.5.11Adverse Events III – CD patients with Other Biologic

| | | | | | ( | Outcome | | |
|---|---|---|---|---|---|---|---|---|
| | Nº pat. (%) | Nº AE | Recovered | Recovering | Not recovered | Recovered with sequelae | Fatal | Unknown |
| <u>Overall</u> | xx (xx.x) | xx | xx | xx | XX | xx | xx | xx |
| SOC 1 | xx (xx.x) | xx | xx | xx | xx | )O) | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx | xx x | xx | XX | XX |
| PT 2 | xx (xx.x) | xx | xx | xx | XX O. | xx | xx | xx |
| | | | | | 0// | | | |
| SOC 2 | xx (xx.x) | xx | xx | XX | US XX | xx | xx | xx |
| PT 1 | xx (xx.x) | xx | xx | xx cic | xx | xx | xx | xx |
| PT 2 | xx (xx.x) | xx | xx | xx (100) | xx | xx | xx | xx |
| | | | | COMI | | | | |
| | | | | 71 | | | | |




Table 5.5.12Adverse Events I – UC patients with VDZ

Table 5.5.13Adverse Events II - UC patients with VDZ

Table 5.5.14Adverse Events III - UC patients with VDZ

Table 5.5.15Adverse Events I – UC patients with Other Biologic

Table 5.5.16Adverse Events II - UC patients with Other Biologic

Table 5.5.17Adverse Events III - UC patients with Other Biologic

All rights reserved. No part of this material may be reproduced or copied in any form by any means (written, electronic, photocopying, recording or otherwise) without the prior consent of BioClever.

SOPs ST 1008-06-II